

# **Face It: Pilot study**

**Evaluation protocol** 

14/09/2023

Alice Worsley, Lilli Wagstaff, Tess Moseley-Roberts, Jack Martin, Tom McBride





# Acknowledgements

We are grateful to colleagues from Khulisa (including Iman Haji and Derellanne Knowles) for their assistance with and input into the early stages of this evaluation. We are also grateful to colleagues from the Behavioural Insights Team (particularly Dr Patrick Taylor, and Leonie Nicks), the Youth Endowment Fund (particularly Dr Mollie Bourne, Dr Daniel Acquah, and Dr Amy Wells) and Dr Nick Axford (University of Plymouth) for their helpful advice and feedback.

We are grateful to the Youth Endowment Fund (originally funded by an endowment from the Home Office) and Stuart Roden for the funding which supports this work, and to the Behavioural Insights Team and Nesta for their support and role in administering this funding.







# **About**

This report was first published in September 2023, and is available to download as a free PDF at: https://www.bi.team/wp-content/uploads/2023/09/Face-It-Pilot-Study-Protocol1.pdf

This work is being undertaken by the Ending Youth Violence Lab at the Behavioural Insights Team. The Behavioural Insights Team (BIT) is a global social purpose company that generates and applies behavioural insights to inform policy, improve public services and deliver results for citizens and society. With company number 08567792.

# **Contents**

| Contents | 2 |
|-----------------------------------------------------------------------|----|
| 1. Study rationale and background | 4 |
| About the Ending Youth Violence Lab | 4 |
| Project overview | 5 |
| 2. Intervention | 6 |
| Intervention overview | 6 |
| Intervention theory of change | 7 |
| How the intervention compares to other services and services-as-usual | 8 |
| 3. Research objectives | 9 |
| 4. Monitoring and success criteria | 12 |
| 5. Design and methodology | 14 |
| Design | 14 |
| Participants | 15 |
| Sample size | 17 |
| Outcome measures | 18 |
| Methods and data collection | 24 |
| Data analysis | 32 |
| Risks to study validity | 33 |
| Qualitative research | 34 |
| 6. Cost evaluation - data collection and reporting | 41 |
| 7. Planned outputs | 42 |
| 8. Ethics and data protection | 42 |
| Ethics | 42 |
| Safeguarding | 44 |
| Data protection | 44 |
| Data management | 45 |
| 9. Racial diversity and inclusion | 47 |
| 10. Risks | 50 |
| 11. Timeline | 52 |
| Annexes | 55 |
| Annex A: Summary of Face It programme using the TIDieR framework | 55 |
| Annex B: Khulisa's Theory of Change narrative and diagram | 62 |
| Annex C: Power calculations | 70 |
| Annex D: Face It milestones | 71 |

| Annex E: Evaluation team experience | 75 |
|------------------------------------------------------------------|----|
| Annex F: Schedule for recruitment, interventions and assessments | 77 |
| Annex G: BIT data protection policy summary | 80 |

| Project title | Face It Evaluation - Pilot study |
|---|---|
| Developer (Institution) | Khulisa |
| Evaluator (Institution) | Ending Youth Violence Lab |
| Principal investigator(s) | Tom McBride |
| Evaluation plan author(s) | Alice Worsley, Lilli Wagstaff, Tess Moseley-Roberts,<br>Jack Martin, Tom McBride |
| Evaluation setting | 5 schools in London |
| Target group | 13-15 year-olds living in London at risk of school exclusion |
| Planned number of participants | 5 schools, approximately 160 young people |
| Funding source and declaration of interests | Funding was received for this work from the Youth Endowment Fund (YEF) and from philanthropist Stuart Roden. There are no known conflicts of interest associated with this publication, and there has been no significant financial support for this work that could have influenced its outcome. |

# 1. Study rationale and background

### About the Ending Youth Violence Lab

The Lab was founded in Summer 2022, bringing together expertise in intervention, evaluation and youth violence. It is funded by Stuart Roden and the Youth Endowment Fund (YEF), and is being incubated at the Behavioural Insights Team (BIT).

The Lab's mission is to catalyse a step change in understanding and tackling violence. To do this, we do 3 things: Firstly, we identify promising projects which seek to address youth violence. Secondly, we fund the development and delivery of those projects. Thirdly, we conduct research to assess how delivery has gone, ways to make it even better, and the potential for further evaluation (with a focus on early-stage testing, to support the work of YEF).

We prioritise three strands of activity:

- Supporting the importation, adaptation, and testing of well-evidenced interventions from overseas - We will identify approaches with strong evidence of improving youth violence outcomes or related upstream factors in other countries, adapt these to the UK context, and deliver early-stage testing.
- Working with UK organisations to develop strong ideas into evaluable interventions - We will work with the sector to find interventions that have strong theoretical underpinnings and are committed to rigorous evaluation, and oversee the development and early-stage testing needed to get them trial-ready.
- 3. Working with developers, researchers, practitioners, and service users to co-design new and innovative approaches - We will build partnerships and fund the development of novel approaches to tackling youth violence, with a focus on addressing underserved populations and unmet needs.

The project described in this protocol forms part of strand 2 of the Lab's approach.

### **Project overview**

Face It is a schools-based intervention, developed by Khulisa. It is an intensive therapeutic group programme for young people, focused on developing social and emotional skills and designed to explore the root causes of emotional distress. It combines creative techniques like storytelling, art, debating, and role-play, using a model informed by neuroscience.

There is strong evidence that social and emotional skills are important for the positive development of children and young people, and contribute to a range of important long-term educational, economic, health, social and criminal justice outcomes<sup>1 2</sup>. There is also good evidence that well-designed school-based social and emotional programmes can be effective, that they are being successfully implemented in UK schools, and can have positive impact on students' social and emotional competencies and educational outcomes<sup>3</sup>.

The Face It intervention is in its early stages in terms of evidence and evaluation, and there is not yet a robust randomised control trial demonstrating that it is effective at improving outcomes for children and young people. However, Face It indicates early promise as an intervention to improve social and emotional skills. The intervention has demonstrated that it can recruit and retain participants, and qualitative work indicates that the programme is well-regarded by participants. An internal evaluation of the programme conducted by Nesta indicated that Khulisa's theory of change highlights relevant outcomes, and both quantitative and qualitative insights suggested largely positive changes in the outcomes examined<sup>4</sup>. Khulisa is also currently conducting a quasi-experimental study which is scheduled to be completed in the Autumn 2023. These studies collectively show that the intervention shows promise.

However, the lack of a randomised comparison group in the existing evaluations limits the conclusions that can be made about impact on outcomes for children and young people. Before any future full-scale randomised control trial, it is important that a small-scale pilot trial is conducted in advance to support and inform this work - to test and improve evaluation procedures such as randomisation and data collection, and to generate useful information around sample size determination.

<sup>&</sup>lt;sup>1</sup> Goodman, A., Joshi, H., Nasim, B., & Tyler, C. (2015). Social and emotional skills in childhood and their long-term effects on adult life.

<sup>&</sup>lt;sup>2</sup> OECD. (2017). Social and emotional skills: Well-being, connectedness and success.

<sup>&</sup>lt;sup>3</sup> Clarke, A. M., Morreale, S., Field, C. A., Hussein, Y., & Barry, M. M. (2015). What works in enhancing social and emotional skills development during childhood and adolescence. A review of the evidence on the effectiveness of school-based and out-of-school programmes in the UK. A report produced by the World Health Organization Collaborating Centre for Health Promotion Research, National University of Ireland Galway.

<sup>&</sup>lt;sup>4</sup> Barber, A. (no date) An internal evaluation of Khulisa's 'Face It' wellbeing programme in schools. rep. Khulisa. Available at:

https://www.khulisa.co.uk/wp-content/uploads/images/NESTA-Evaluation-Report-2020.pdf.

# 2. Intervention

#### Intervention overview

This project is a pilot evaluation of Face It, a school-based intervention designed and implemented by Khulisa. Face It is specifically designed for young people at risk of offending, exploitation, and school exclusion. The programme builds self-awareness and encourages pupils to reflect on the root causes and triggers of their disruptive or challenging behaviour. Khulisa believes that early intervention breaks the school to prison pipeline, which is exacerbated by exclusion, enabling young people to choose a safe and crime-free future. The intervention is delivered over 6 weeks, including an intensive 5-day programme of activities, and pre-programme and post-programme group and 1:1 sessions. Each programme is tailored to participants' needs and uses art, storytelling, 1:1 and group experiential techniques, delivered by trained dramatherapists. Programme facilitators are assigned to groups of young people ensuring that at least one person on each facilitation team has a therapeutic qualification. This is typically a dramatherapy qualification, but may also be relational therapy. A detailed description of Face It using the TIDieR framework can be found in Annex A.

Face It aims to help young people learn new coping mechanisms and skills to identify individual triggers (for example anger, conflict etc.) and alternative responses that can help improve capacity for concentration and focus during lessons. It has a focus on developing emotional regulation skills (planning, decision making, and communication) which can have a positive impact on behaviour, sense of self-worth and confidence.

Figure 1 details a high level Theory of Change for the intervention. A logic model developed by Khulisa can be found in Annex B. We have conducted an initial review of the Theory of Change and discussed this in depth with Khulisa and have concluded that the outcomes they specify and the underlying pathways to achieve them are sufficiently well considered and plausible to justify further evaluation.

### Intervention theory of change



Figure 1 - Face It theory of change

### How the intervention compares to other services and services-as-usual

Face It can be distinguished from many other school-based social and emotional programmes for similar cohorts on the basis that it is delivered by therapeutically qualified practitioners and combines 1:1 sessions with group sessions. In particular:

- It takes a therapeutic and trauma-informed approach: Khulisa's programmes are led by therapists and follow trauma-informed methodologies including Perry's neurosequential model<sup>5</sup> <sup>6</sup>.
- 2. Its activities are creative and experiential: It is theorised that children with limited emotional literacy respond more effectively to non-verbal activities. Khulisa uses art, drama therapy, role play and games to help participants observe themselves through the experiences of others, which is intended to help them understand the behaviours that benefit or hold them back.
- **3.** The programme combines group and 1:1 support to embed learning: Face It uses a multi-layered approach to learning. 1:1 sessions give facilitators an opportunity to get an insight into participants' levels of self-awareness and shed light on how to help these participants build confidence, self-worth, and more positive and healthy beliefs. Group sessions aim to enable participants to build relationships, develop empathy and learn to respect other perspectives through group discussion, and other activities.

<sup>&</sup>lt;sup>5</sup> Perry, B.D (2006) 'Applying principles of neurodevelopment to clinical work with maltreated and traumatized children: the Neurosequential Model of Therapeutics' in Webb, N.B (Eds.) *Traumatized youth in child welfare*, Guildford Press, New York, 27 – 51.

<sup>&</sup>lt;sup>6</sup> Perry, B.D (2009) Examining child maltreatment through a neurodevelopmental lens: clinical applications of the Neurosequential Model of Therapeutics, *Journal of Loss and Trauma*, 14, 240 – 255.

# 3. Research objectives

This pilot trial is not primarily designed to estimate effect sizes or evaluate the impact of the intervention, but is instead focused on **assessing if Face It could and should progress to more rigorous evaluation**. If the pilot trial is successful (based on the criteria discussed in *Section 3*), then there is a strong case for this to progress to a full-scale efficacy trial to examine impact across a range of outcomes. Ideally this future evaluation would be adequately powered to adjust for multiple comparisons, explore moderating and mediating factors, and analyse differential impacts on pre-specified subgroups.

The pilot trial is designed to test the following questions:

- **Feasibility** Can Face It recruit and retain sufficient numbers of young people from the target population, and be delivered with fidelity?
- Acceptability Do young people value the programme and feel that the content and delivery are appropriate to their needs? Do teachers and caregivers find programme delivery acceptable?
- Evaluability Do we have enough confidence in the feasibility of a randomised controlled trial (RCT), particularly in terms of recruitment into evaluation, randomisation and outcome data collection, to justify a future full-scale efficacy trial?
- Outcomes Does Face It show sufficient promise in terms of improvements in key outcomes (resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions) to justify a subsequent efficacy trial?<sup>7</sup>
- Mechanisms Is it possible to collect data which would allow for the testing of mediators, moderators and differential impact as part of any subsequent evaluation?

More detail on how we will address these questions is provided in *Table 1*.

<sup>&</sup>lt;sup>7</sup> Note that the sample size in this pilot is unlikely to be big enough to make strong causal claims about effectiveness. However, it should be sufficient for us to produce descriptive statistics on key outcome variables and make an estimate of effectiveness with low levels of confidence.

Table 1 Research questions

| Tubic | Research questions | |
|---|---|---|
| | Overarching Question | Sub-question |
| Feasibility | Can Face It recruit and retain sufficient numbers of young people from the target population, and be delivered with fidelity? | <ul> <li>Reach and recruitment</li> <li>Can Khulisa recruit a sufficient number of schools to participate in the programme?</li> <li>Can Khulisa recruit and retain sufficient young people at risk of youth violence?</li> <li>What factors affect recruitment and retention?</li> <li>Do recruitment and retention vary by ethnicity, gender or other baseline characteristics?</li> <li>How should the programme be adapted to improve recruitment and retention?</li> <li>Fidelity</li> <li>Can Face It be delivered with fidelity?</li> <li>What factors affect fidelity?</li> <li>What variations in delivery are appropriate for effective implementation?</li> </ul> |
| Acceptability | Do young people value the programme and feel the content and delivery are appropriate to their needs? Do teachers and caregivers find programme delivery acceptable? | <ul> <li>Is Face It acceptable to young people at risk of youth violence?</li> <li>Does participation in a randomised evaluation affect participants' views of the intervention? If so, how?</li> <li>Does acceptability vary by ethnicity and race?</li> <li>Is the programme acceptable to schools?</li> <li>What factors affect acceptability?</li> <li>How could the programme be adapted to increase acceptability?</li> </ul> |
| Evaluability | Do we have enough confidence in the feasibility of a randomised controlled trial, particularly in terms of recruitment into evaluation, randomisation and outcome data collection, to justify a continuation of the efficacy trial? | <ul> <li>Is randomisation feasible and adhered to?</li> <li>Is data collection possible and sufficient?</li> <li>What factors affect ease of data collection and completeness and quality of data?</li> <li>How could the approach to data collection be improved to increase ease, completeness and quality?</li> <li>Is it possible to retain schools and young people in the control group?</li> <li>What factors affect retention in the control group? What are the best methods of achieving retention in the control group?</li> <li>Do practitioners or young people feel that the evaluation impacts on intervention delivery? If so, what elements of the intervention affect delivery quality?</li> <li>Is randomisation acceptable to practitioners &amp; teachers?</li> <li>What factors affect acceptability?</li> </ul> |

| | | How could the approach to randomisation be adapted to increase acceptability? |
|---|---|---|
| Outcomes | Does Face It show sufficient promise in terms of improvements in key outcomes to justify a subsequent efficacy trial? | Is there preliminary evidence that Face It improves: |
| Mechanisms<br>and<br>moderating<br>factors | Is it possible to collect data which would allow for the testing of mediators and moderators and differential impact as part of any subsequent YEF evaluation? | <ul> <li>Is it possible to gather data and permissions so that a future RCT could assess:</li> <li>If outcomes vary by: <ul> <li>School type or location</li> <li>Gender</li> <li>Age</li> <li>SES/FSM</li> <li>Race and ethnicity</li> </ul> </li> <li>Which part of Face It leads to improved outcomes?</li> </ul> |

# 4. Monitoring and success criteria

We will use Pause/Go criteria for two purposes:

- 1. Throughout the evaluation to monitor if the pilot is proceeding as expected, allowing for us to make real time adjustments or pause the work if needed. Criteria scoring in red or amber zones will prompt changes to the pilot trial process, and, if criteria do not improve, may prompt termination of the trial.
- 2. At the end of the evaluation to make recommendations to YEF as to whether a full RCT should be pursued.

Criteria used to monitor ongoing trial progress are as follows:

1) Recruitment I: Number of schools successfully recruited to the evaluation in the first 3 months of the pilot (addresses feasibility and evaluability)

a) Red: 3 or fewer

b) Amber: 4

c) Green: 5

2) Recruitment II: Proportion of target number of eligible young people recruited within schools in the first 3 months of the pilot<sup>8</sup> (addresses **feasibility**)

a) Red: <60% of target</li>

b) Amber: 60-79% of target c) Green: 80-100% of target

3) Randomisation: Proportion of recruited young people randomised to control or treatment groups (addresses feasibility, evaluability and acceptability)

a) Red: <50%

b) Amber: 50-79%

c) Green: 80-100%

4) Retention: Proportion of young people in the intervention arm completing the intervention<sup>9</sup> (addresses feasibility and acceptability)

a) Red: <50%

b) Amber: 50-79%

- c) Green: 80-100%
- 5) Fidelity: Assessed by the Lab through comparing facilitator self-report of activities conducted during the 5-day programme with Face It's list of key activities, found in Annex D, which was developed in collaboration with the delivery team prior to the pilot study (addresses feasibility)

<sup>8</sup> Assuming delivery in two cohorts over two school terms with a 3-month follow up for the first cohort only, we anticipate that the trial will last approximately 6-7 months

Defined as attending both pre-programme and post-programme group and 1:1 sessions and all 5 days of the delivery

a) Red: <50% of sessions meet at least 80% of criteria

b) Amber: 50-79% of sessions meet 80% of criteria

c) Green: 80-100% of sessions meet 80% of criteria

Criteria used to contribute to determining recommendations to YEF are as follows:

1) Outcomes I: Data completeness for YP self-reported outcome variables post intervention<sup>10</sup> for treatment and control (addresses **evaluability**)

a) Red: <35%</li>
 b) Amber: 35-89%
 c) Green: 90-100%<sup>11</sup>

2) Outcomes II: Data completeness for YP self-reported outcome variables at 3 months post intervention for treatment and control (addresses **evaluability**)

a) Red: <35%</li>b) Amber: 35-89%c) Green: 90-100%

- 3) Outcomes III: Directional change in outcome variables for treatment and control (addresses **outcomes**)
  - a) Red: at least one outcome measure indicates negative results and no positive results 12
  - b) Amber: null or mixed results
  - c) Green: at least one outcome measure indicates positive results and no negative results

Monitoring criteria will focus primarily on data completeness for young people, as our primary outcome measure is the self-reported SDQ at post-programme. We will also monitor response rates of parent surveys, although without specified thresholds. This will inform our reporting to YEF, such as whether a full scale trial should incorporate parent-reported metrics, and how best to approach this.

We will also record response rates for the 3-month follow up survey for young people. As delivery will take place in two cohorts, one in the Autumn term and one in the Spring term, the timeline for 3-month follow-up for the Spring term delivery cohort will fall towards the end of the academic year. As such, we anticipate that response rates for this cohort may be lower. Again, we will monitor this without stringent thresholds in order to inform recommendations about the timing of delivery and data collection.

<sup>&</sup>lt;sup>10</sup> We will have 100% completion for pre-test by definition, as students are not eligible for randomisation if they did not complete pre-test assessment measures

<sup>&</sup>lt;sup>11</sup> Thresholds based on the EIF evidence standards guidelines (available at: https://guidebook.eif.org.uk/eif-evidence-standards)

<sup>&</sup>lt;sup>12</sup> Null results: 95% confidence intervals that cross 0; negative results: 95% confidence intervals that are entirely below 0; positive results: 95% confidence intervals that are entirely above 0

# 5. Design and methodology

# Design

This pilot trial will be a parallel two-armed randomised controlled superiority trial of Face It compared to services as usual (SAU) for young people at risk of exploitation, offending and school exclusion. The unit of randomisation will be individual pupils. A pragmatic sample of state secondary schools in areas with high levels of violence in England (e.g. located in a Violence Reduction Unit) will be selected. We will aim to recruit schools with a high proportion of disadvantaged pupils (more pupils in receipt of the Pupil Premium than the national average) and that are ethnically diverse (at least 30 per cent of pupils not of white British heritage). This will not be a waitlist control study, as this pilot study is designed to assess the feasibility of a full-scale efficacy trial including offending as an outcome. This requires long-term follow-up, hence a waitlist would not be possible. This may affect recruitment and retention of schools in the study, as this design will mean that many eligible pupils will not receive the intervention, and schools will have no control over which students receive the programme. However, we will work with Khulisa to mitigate this risk by emphasising the importance of the trial to schools and participants, encouraging attendance at data collection activities through food incentives, and ensuring that the process is simple and straightforward for participants to minimise friction.

The pilot trial will use a within-schools randomisation design, with randomisation taking place at the level of the individual student. Baseline assessment will be conducted by researchers who are blind to treatment allocation as young people will not yet have been allocated to control or intervention groups. We will endeavour to blind the researcher conducting post-treatment data collection by ensuring that data collection is arranged by a different researcher. This means that the researcher will not have been involved in the scheduling, and will not know who is in their session and their treatment allocation. However, it is possible that young people may ask questions of the evaluator, such as seeking clarification on survey questions, that may indicate their allocation. Young people, teachers and families are not blind to treatment allocation.

We will attempt to recruit an overall sample with an approximately 80:20 split of participants displaying primarily externalising and internalising behaviours respectively, as Khulisa views this balance as an essential component of building an optimal group dynamic for the programme. We will then use stratified randomisation to ensure that participants within the treatment group and control group are balanced on these characteristics and the 80:20 split is maintained in each. Pupils will be classified into groups with internalising or externalising behaviour based on the referral form completed by schools. We will also stratify by gender to ensure the treatment and control group are balanced on this characteristic - and particularly so that there is a sufficient balance within the treatment group to facilitate mixed-gender intervention groups, which the programme developers argue improves group dynamics.

If schools refer a number of young people that exceeds the desired sample size (as discussed below), we will conduct a two stage randomisation process. First, we will randomly select a subsample of the referred students, limited to the maximum sample size per school. Second, we will randomly assign members of this subsample to either treatment or control. Those not randomly selected will not participate in the programme or the study. This will ensure that we do not over sample in either the treatment or control group and that allocation to the treatment group is entirely random.

Randomisation and assignment to intervention or control groups will be implemented by the Ending Youth Violence Lab using a random number generator in Stata. The allocation mechanism will be young people's Unique Pupil Number (UPN).

Randomisation will occur in batches for each school after students are referred to the programme and assessed for eligibility, and after consent has been obtained and baseline assessment has taken place, but before any contact with the programme such as 1:1 discussions. This means that after Khulisa has received referrals and assessed eligibility, the Ending Youth Violence Lab will conduct baseline data collection and randomise eligible students to either treatment or control on a 1:1 ratio in each school in turn. The Ending Youth Violence Lab will then inform Khulisa about the allocation of young people to treatment or control.

Individuals allocated to the control group will receive services as usual (SAU). As part of data collection, we will investigate what this entails through surveys of control group participants.

As part of the development of this pilot study, we will conduct a participatory panel with a separate group of young people who have experienced the programme in the past few years. We will seek input from the panel on the design of our evaluation materials and in interpreting our findings.

# **Participants**

Participants will be young people aged 13-15 in years 9 and 10, who are referred to Face It by schools and who meet programme eligibility criteria. Referrals will be made within-school, typically by teachers with awareness of the pupil's behaviour, such as a Head of Year or Form Tutor, and based on recruitment criteria shared with schools by Khulisa. Pupils will be identified as at risk due to internal school data and assessed for eligibility using information from Khulisa's referral form. Participants will then be enrolled by Khulisa.

The programme will be delivered within 5 schools, twice within each school, to two different groups of young people (to one group of Year 9s, and to one group of Year 10s).

Participants will predominantly be pupils displaying externalising behaviours. This indicates pupils at risk of youth violence, proxied by risk of exclusion, history of verbal or physical violence and/or bullying perpetration. Participants will also include pupils displaying

internalising behaviours. This includes young people with low self esteem and at risk of bullying victimisation. Programme groups will include young people displaying externalising and internalising behaviours with an approximate ratio of 80:20 as Khulisa views this balance as an essential component of building a group dynamic.

All participants will be asked to consent to be part of the evaluation for ethical purposes before data collection and randomisation. We will seek consent for participation in the evaluation first from the Head Teacher or other member of the senior leadership team who is capable of acting *in loco parentis*. This individual will provide written consent for pupils within the school to participate in the evaluation and receive the programme.

Parents/caregivers of young people will be given an information sheet explaining the evaluation purpose and process and will be given the opportunity to withdraw their child from the evaluation. Young people will be given a verbal explanation of the purpose and process of the evaluation as well as a written information sheet. Young people will be asked for active written consent prior to survey data collection, and will be given the opportunity to opt out of data processing of routinely collected school data. Participation in the intervention is contingent on participation in the evaluation, hence opting out of data collection prior to intervention delivery would involve withdrawing from the programme. Young people will also have the opportunity to opt out of data processing and/or the evaluation at a later stage by speaking to a teacher.

Young people will also be asked for written consent in order to participate in interviews.

The same pathway for consent as detailed above will be applied for participation in the participatory panel: the Head Teacher, or other appropriate staff member, will consent for the school to participate. Parents/caregivers of young people will then be given the opportunity to withdraw their child, and young people will give written consent to participate.

Participating schools will be identified by Khulisa using convenience sampling. The limitations of this approach will be highlighted in the final report. All schools identified will be in London. Individual recruitment will take place following Face It's usual processes with the additions of explanations of the trial and randomisation.

Figure 2 below outlines the proposed participant flow for the project.



Figure 2 - Participant flow diagram for pilot study

# Sample size

Khulisa has significant experience delivering Face It and has determined that the ideal group size is between 8-10 students. Through our discussion with them, it became clear that

recruiting more than 5 schools would not be feasible in the timelines of the pilot. However, they are able to deliver the programme to two cohorts of students in each school. We therefore will aim to recruit 160 eligible participants across five schools (80 young people in the intervention group and 80 in the control group). Khulisa will ask schools to refer anyone who is eligible for the intervention. This will give us a stronger understanding of the true demand for interventions like Face It in schools.

We will use a pragmatic approach to achieve an overall sample size of 160 eligible participants: if some schools are unable to refer a sufficient number of pupils, we will aim to oversample from other schools, noting that Khulisa can deliver the programme in groups of up to 12.

Using pupil level randomisation, a sample size of 160, power of 0.8, and estimates for standard deviation on the SDQ from previous papers<sup>13</sup>, we anticipate that we would be able to detect a Cohen's D of 0.5 (or a mean difference of 3 on the SDQ). Whilst this effect size is larger than those detected in many YEF efficacy trials (or used in the power calculations), our primary objective in this study is not to test the impact of Face It, but rather to establish its evaluability and generate information that will enable a full-scale impact evaluation in the future.

It is worth noting that during this pilot trial we are making no assumptions about pre-test post-test correlation, which means our power calculations are conservative estimates. As part of this study we aim to collect sufficient data to make an estimate of this value (and the standard deviation of the outcome) to enable more accurate power calculations for any full-scale efficacy trial.

### Outcome measures

We intend to have one primary outcome (the self-assessment Strengths and Difficulties Questionnaire at post-programme), and a number of secondary outcomes. Given the high number of outcomes and comparisons we will be making, we will be adjusting for multiple comparisons. While this is not strictly necessary in a pilot study where the aim of the trial is not to estimate impact, we feel it is important to replicate the analytical approach which would be used in a full scale efficacy trial. More details on how we will adjust for multiple comparisons can be found in the Statistical Analysis Plan. All outcome measures (see Table 2) will be collected at baseline (prior to the intervention), at post-test (after delivery of the intervention), and at 3-month follow-up (with the exception of attendance and exclusions, which will only be collected at baseline and follow-up).

<sup>&</sup>lt;sup>13</sup> Two papers found that the standard deviation for the SDQ was between 5-7, so we ran our power calculations assuming 6.5. The papers are cited as follows: Cortina, Melissa & Fazel, Mina. (2014). The Art Room: An Evaluation Of A Targeted School-based Group Intervention For Students With Emotional And Behavioural Difficulties.. The Arts in Psychotherapy. 11. 10.1016/j.aip.2014.12.003; Vugteveen, J., de Bildt, A. & Timmerman, M.E. Normative data for the self-reported and parent-reported Strengths and Difficulties Questionnaire (SDQ) for ages 12–17. Child Adolesc Psychiatry Ment Health 16, 5 (2022). https://doi.org/10.1186/s13034-021-00437-8

Table 2 Outcome measures

| Type of outcome | Outcome<br>measured | Instrument | Completed<br>by | Number<br>of items | Age<br>suitability<br>(young<br>person) | Subscales to be used | Scoring <sup>14</sup> | References |
|---|---|---|---|---|---|---|---|---|
| Primary | Behavioural difficulties | Strengths and Difficulties Questionnaire (SDQ) - post-programme self-assessment | Young person | 25 | 11-17 | All subscales including: Emotional symptoms Conduct problems Hyperactivity/inattention Peer relationships problems Prosocial behaviour | Total difficulties score: A score from 0-40 is generated by summing scores from all the subscales, except the prosocial subscale. While the total difficulties score is the primary outcome, we will also examine the total difficulties score when broken down into the externalising score (the sum of the conduct and hyperactivity scales), and the internalising score (the sum of the emotional and peer problems scales). | Goodman,1997 <sup>15</sup> |

Data will be collected and outcome measures scored by the Ending Youth Violence Lab
 Goodman R (1997) The Strengths and Difficulties Questionnaire: A Research Note. Journal of Child Psychology and Psychiatry, 38, 581-586.

| Secondary | Behavioural<br>difficulties | SDQ - 3-month follow-up self-assessment | Young<br>person | 25 | 11-17 | <ul> <li>All subscales including:</li> <li>Emotional symptoms</li> <li>Conduct problems</li> <li>Hyperactivity/inattention</li> <li>Peer relationships problems</li> <li>Prosocial behaviour</li> </ul> | Total difficulties score: A score from 0-40 is generated by summing scores from all the subscales, except the prosocial subscale. Summed score of subscales give a score ranging from 0-40s | Goodman,1997 <sup>16</sup> |
|---|---|---|---|---|---|---|---|---|
| | Behavioural<br>difficulties | SDQ - parent assessment | Parent/care giver | 25 | 4-17 | <ul> <li>All subscales including:</li> <li>Emotional symptoms</li> <li>Conduct problems</li> <li>Hyperactivity/inattention</li> <li>Peer relationships problems</li> <li>Prosocial behaviour</li> </ul> | Total difficulties score: A score from 0-40 is generated by summing scores from all the subscales, except the prosocial subscale. | Goodman,1997 <sup>17</sup> |
| | Offending | The Self-Report<br>Delinquency<br>Scale | Young<br>person | 19 | 10-17 | Does not have subscales | Variety of delinquency score: Sum the number of items the respondent answers 'yes' to: • Yes = 1 • No = 0 Produces a score that | Thornberry and Krohn, 2000 <sup>18</sup> |

<sup>&</sup>lt;sup>16</sup> Goodman R (1997) The Strengths and Difficulties Questionnaire: A Research Note. Journal of Child Psychology and Psychiatry, 38, 581-586. <sup>17</sup> Goodman R (1997) The Strengths and Difficulties Questionnaire: A Research Note. Journal of Child Psychology and Psychiatry, 38, 581-586.

<sup>&</sup>lt;sup>18</sup> Thornberry, T.P., & Krohn, M.D. (2000). The self-report method for measuring delinquency and crime. Measurement and Analysis of Crime and Justice, 4, 33-83.

21

| | | | | | | ranges from 0-19. Volume of delinquency score: Summing the point values when respondents report a number of times. Point values are assigned as follows: • Once = 1 • Twice = 2 • 3 times = 3 • 4 times = 4 • 5 times = 5 • Between 6 and 10 times = 6 • More than 10 times = 11 | |
|---|---|---|---|---|---|---|---|
| Victimisatio<br>n | Problem<br>Behaviour<br>Frequency Scale | Young person | 10 | Adolescents | <ul><li>Overt victimisation</li><li>Relational victimisation</li></ul> | A score ranging from<br>6-36 achieved by<br>summing scores of the<br>two subscales | Farrell et al., 2016 <sup>19</sup> |
| Resilience | Children's Hope<br>Scale | Young<br>person | 6 | 8-16 | All subscales | A score ranging from<br>6-36 achieved by<br>summing scores of the | Snyder et al.,<br>1997 <sup>20</sup> |

<sup>&</sup>lt;sup>19</sup>Farrell, A. D., Sullivan, T. N., Goncy, E. A., & Le, A. T. H. (2016). Assessment of adolescents' victimization, aggression, and problem behaviors: Evaluation of the Problem Behavior Frequency Scale. *Psychological assessment*, 28(6), 702.

<sup>&</sup>lt;sup>20</sup> Snyder, C. R., Hoza, B., Pelham, W. E., Rapoff, M., Ware, L., Danovsky, M., ... & Stahl, K. J., "The development and validation of the Children's Hope Scale," *Journal of Pediatric Psychology*, Vol. 22, No. 3, 1997, pp. 399–421.

| | | | | | | two subscales | |
|---|---|---|---|---|---|---|---|
| Emotional regulation | The Emotional<br>Regulation<br>Questionnaire | Young<br>person | 10 | 10-18 | <ul> <li>Cognitive reappraisal</li> <li>Expressive suppression</li> </ul> | Summed score of subscales. The higher the score, the greater the use of emotion regulation strategies, conversely lower scores represent less frequent use of such strategies | loannidis & Siegling, 2015 <sup>21</sup> Gross & John, 2003 <sup>22</sup> Gullone & Taffe, 2012 <sup>23</sup> |
| Social and emotional wellbeing | The Short<br>Warwick-Edinbur<br>gh Mental<br>Well-being Scale<br>(SWEMWBS) | Young person | 7 | 11+ | Does not have subscales | The SWEMWBS is scored by first summing the scores for each of the seven items, which are scored from 1 to 5. The total raw scores are then transformed into metric scores using the SWEMWBS conversion table resulting in a score ranging from 7-35. | Melendez-Torres et al., 2019 <sup>24</sup> |

<sup>&</sup>lt;sup>21</sup> loannidis, C. A., & Siegling, A. B. (2015). Criterion and incremental validity of the emotion regulation questionnaire. Frontiers in Psychology, 6, Article 247. https://doi.org/10.3389/fpsyg.2015.00247 <sup>22</sup> Gross, J.J., & John, O.P. (2003). Individual differences in two emotion regulation processes: Implications for affect, relationships, and well-being. Journal of Personality and Social Psychology, 85, 348-362.

<sup>&</sup>lt;sup>23</sup> Gullone, Eleonora; Taffe, John (2012). The Emotion Regulation Questionnaire for Children and Adolescents (ERQ–CA): A psychometric evaluation.. Psychological Assessment, 24(2), 409–417. doi:10.1037/a0025777

<sup>&</sup>lt;sup>24</sup>Melendez-Torres, G., Hewitt, G., Hallingberg, B. et al. Measurement invariance properties and external construct validity of the short Warwick-Edinburgh mental wellbeing scale in a large national sample of secondary school students in Wales. Health Qual Life Outcomes 17, 139 (2019). https://doi.org/10.1186/s12955-019-1204-z

| School attendance | ImpactEd data | Admin data | N/A | N/A | N/A | Number of absences during the pilot period | N/A |
|---|---|---|---|---|---|---|---|
| School exclusions | ImpactEd data | Admin data | N/A | N/A | N/A | Number of exclusions during the pilot period | N/A |

Additionally, while a subsequent efficacy trial will evaluate violence as an outcome, it will not be measured in this pilot trial due to the short timeframes: data from Police National Computer (PNC) records, which represent the most reliable data, will not be available for several years. We will, however, test that we can collect data and obtain consent (for ethical reasons) for analysis of PNC data to provide assurance to YEF that analysis of the impact on offending would be feasible in any subsequent efficacy trial. We will also collect self-reported offending data from young people using the Self-Report Delinquency Scale.

#### Methods and data collection

#### Quantitative research activities

We will be conducting quantitative research activities within all five participating schools. We will use:

- a) Young person survey at baseline, end-of-programme and 3-months post-programme
- b) Parent/caregiver survey at baseline, end-of-programme and 3-months post-programme
- c) Programme administrative data
- d) ImpactEd data
- e) Facilitator report

#### a) Young person survey

We will conduct surveys with young people at baseline (pre-randomisation), end-of-programme and at 3-months post-programme. Surveys will be conducted in person in groups during the school day. Since all outcome measures we have chosen can be self-administered, young people will complete the survey themselves using technology provided by schools such as computers or tablets. However, to ensure the data that is collected is of high quality, a trained member of the evaluation team will be present at all data collection sessions to respond to any clarification questions. To ensure the conditions are as similar as possible across all data collection sessions, Lab staff will be trained on how to facilitate these sessions, highlighting what questions from participants they can answer and what questions they can't. While online completion reduces the likelihood of encountering certain issues relative to paper completion (e.g. errors with digitisation), there will still be opportunities for errors, e.g. participants accidentally skipping questions. We have decided not to make questions mandatory - this is because giving participants the chance to not answer questions that they do not want to was highlighted as a key part of making the survey ethical and fair for participants. To mitigate the potential for accidental skipping of questions, we have included a reminder at the bottom and top of each survey page for participants to check each page is complete before submitting. In addition, Lab staff will remind participants before they begin the survey and before they submit it. Another advantage to online surveys is that we can track the time-to-completion. For details on how we will use this to understand data quality, please see the Statistical Analysis Plan.

We have decided to collect survey data from control and intervention participants separately, as part of separate data collection sessions, rather than collecting survey data from all participants as part of the same groups in the same data collection sessions. There are pros and cons to each of these approaches. On balance, we have opted for the former as our partners at Khulisa felt that the latter would not be feasible, and that it would cause potential issues for the control group to interact with pupils who have received the programme in this context. From an evaluation perspective, there are associated risks around resentful demoralisation and compensatory rivalry.

As the surveys are self-completed by participants, there is arguably limited potential for bias introduced by researchers not being blind to treatment allocation. However, we will endeavour to blind the independent researcher supervising survey completion to treatment allocation by ensuring that data collection is arranged by a different researcher. This means that the researcher will not have been involved in the scheduling, and will not know who is in their session and their treatment allocation. However, it is possible that young people may ask questions of the evaluator, such as seeking clarification on survey questions, that may indicate their allocation.

Each survey collection session will start with a short icebreaker activity. The aim of this activity is to ensure that young people are comfortable in the setting prior to any data collection activities in order to minimise any potential distress from survey questions regarding delinquency, emotional regulation and wellbeing which may be distressing for young people.

#### b) Parent/caregiver survey

We will conduct surveys with parents/caregivers of young people at baseline (pre-randomisation), end-of-programme, and at 3-months post-programme. Surveys will be completed online: parents/caregivers will receive a link to complete the survey via email. Parents/caregivers will be offered a shopping voucher as an incentive to participate.

Since this survey will be completed independently without a trained researcher, the steps we can take to ensure data quality are limited. However, we will inform participants at the beginning of the survey about what the ideal conditions will be. Additionally, we will include reminders at the top and bottom of each page reminding them to check the page is complete before moving on. Finally, we will use the time-to-completion as a check for data quality.

#### c) Programme administrative data

Khulisa will send referral data from referral forms and session attendance lists to the Ending Youth Violence Lab. Programme data will also be recorded and shared, including:

- Number of young people referred;
- Number of eligible participants consenting to participate in the intervention and evaluation:
- Number of young people in the intervention and control arms; and
- Complaints submitted to Khulisa and school staff.

#### d) ImpactEd data

We will use the ImpactEd platform to record school attendance and exclusions. This will be collected at baseline and 3-months post-programme, and linked to participant data using young people's UPNs.

#### e) Facilitator report

Programme facilitators will report activities conducted during the 5-day programme. This will be compared to the Face It milestones (Annex D) to assess programme fidelity (dose and adherence).

Table 3 provides an overview of our proposed methods of data collection. Further detail can be found below. Information on the timings of data collection can be found in Annex F.

Table 3 Data collection - brief overview

| Purpose | Topic | Method <sup>25</sup> | Data collected | Data analysis |
|---|---|---|---|---|
| Feasibility | | Programme administrative data | Number of eligible young people agreeing to intervention and participating in the evaluation | Descriptive statistics |
| | Recruitment | In depth interviews with key school staff who manage relationship with Khulisa: one interview per case study school <sup>26</sup> | Perception of ease of recruiting eligible young people | Framework analysis |
| | | Written reflection from Khulisa on the process of school recruitment including the number of schools approached and how schools were successfully approached | Number of schools approached, successfully engaged and recruited | Descriptive statistics and/or framework analysis |
| | Retention | Programme administrative data | <ul> <li>Number of young people in the intervention arm completing the intervention and completing data collection</li> <li>Number of young people in the control completing the data collection</li> </ul> | Descriptive statistics |
| | Fidelity | Facilitator report | Programme facilitator data on activities delivered compared to Face It milestones <sup>27</sup> - examines dose and adherence | Descriptive statistics |

Orange: quantitative data; Blue: qualitative data; Green: quantitative and/or qualitative See Qualitative Research section for more details

<sup>&</sup>lt;sup>27</sup> Annex D

| | | Interviews with young people | Discussion of young person engagement with programme - examines engagement | Framework analysis |
|---|---|---|---|---|
| | | In-depth interview with one programme facilitator per case study school (between 1 - 3 depending on whether facilitator runs session in more than 1 school) | Details on activities delivered and comparisons to ethos of delivery and experiences running the programme - examines adherence, engagement and quality of delivery | Framework analysis |
| | | Programme administrative data | Compliance with randomisation measured via attendance sheets | Descriptive statistics |
| | Acceptability of randomisation | Programme administrative data | Complaints submitted to Khulisa and school staff | Descriptive statistics |
| | | Programme administrative data | Content analysis of complaints filed | Framework analysis |
| Acceptability | Acceptability of content | Young person post-programme survey | Responses to questions measuring experiences in the intervention | Descriptive statistics |
| | | Interviews with 4-6 young people per school across three schools | Young people's perception of the quality of the content and delivery of Face It | Framework analysis |
| | Acceptability of delivery | In depth interviews with key school staff who manage relationship with Khulisa: one interview per case study school | School staff acceptance of programme | Framework analysis |
| | Completeness of data collection | Young person baseline, post-programme and 3-month post-programme follow-up survey | Admin data on completion of outcome measures from treatment and control | Descriptive statistics |
| Evaluability | Service as usual | Young person post-programme survey | Control group responses about services received | Descriptive statistics |
| | Feasibility of | Short parent/caregiver interviews held at a drop in | Engagement rates for interviews with | Descriptive statistics |

| | interviewing caregivers | evening at one case study school | parents/caregivers within one case study school | |
|---|---|---|---|---|
| | Feasibility of<br>linking to<br>Metropolitan<br>Police dataset | Discussion with Metropolitan police and/or other relevant departments and agencies | Discussion about the feasibility of linking data to the Police National Computer (PNC) | Reporting of outcomes of discussion |
| Outcomes | Resilience | Young person baseline, end-of-programme and 3-month post-programme follow-up survey | The Children's Hope Scale | Pre-specified statistical analysis <sup>28</sup> |
| | | Interviews with young people | Perceptions of behaviour change related to resilience | Framework analysis |
| | | Short parent/caregiver interviews held at a drop in evening at one case study school | Perceptions of behaviour change related to resilience | Framework analysis |
| | Emotional<br>regulation | Young person baseline, end-of-programme and 3-month post-programme follow-up survey | The Emotional Regulation Questionnaire | Pre-specified statistical analysis |
| | | Interviews with young people | Perceptions of behaviour change related to emotional regulation | Framework analysis |
| | | Short parent/caregiver interviews held at a drop in evening at one case study school | Perceptions of behaviour change related to emotional regulation | Framework analysis |
| | Social and emotional wellbeing | Young person baseline, end-of-programme and 3-month post-programme follow-up survey | Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) | Pre-specified statistical analysis |
| | | Interviews with young people | Perceptions of behaviour change related to social and emotional wellbeing | Framework analysis |

<sup>&</sup>lt;sup>28</sup> See Data Analysis section for more details

| | | Short parent/caregiver interviews held at a drop in evening at one case study school | Perceptions of behaviour change related to social and emotional wellbeing | Framework analysis |
|---|---|---|---|---|
| | Behavioural<br>difficulties | Young person baseline, end-of-programme and 3-month post-programme follow-up survey | SDQ (self assessment) | Pre-specified statistical analysis |
| | | Caregiver baseline, end-of-programme and 3-month post-programme follow-up survey | SDQ (parent assessment) | Pre-specified statistical analysis |
| | | Interviews with young people | Perceptions of behaviour change related to behavioural difficulties | Framework analysis |
| | | Short parent/caregiver interviews held at a drop in evening at one case study school | Perceptions of behaviour change related to behavioural difficulties | Framework analysis |
| | Offending | Young person baseline, end-of-programme and 3-month post-programme follow-up survey | Self-report delinquency scale | Pre-specified statistical analysis |
| | Victimisation | Young person baseline, end-of-programme and 3-month post-programme follow-up survey | Problem Behaviour Frequency Scale (overt and relational victimisation subscales only) | Pre-specified statistical analysis |
| | Attendance | ImpactEd data collected at baseline and 3-months post-programme | Attendance data | Pre-specified statistical analysis |
| | Exclusions | ImpactEd data collected at baseline and 3-months post-programme | Exclusion data | Pre-specified statistical analysis |
| Mechanisms | Individual<br>demographics | Programme administrative data (via referral forms) | Data on completeness of data provided | Descriptive statistics |
| | Intervention | Facilitator report | Analysis of the completeness of responses to the Face It Milestones | Descriptive statistics |
| | Feasibility of | Interviews with young people | Analysis of sign-up rates and attendance at | Descriptive statistics |

| conducting<br>interviews | | interviews | |
|---|---|---|---|
| | Interviews with key school staff who manage relationship with Khulisa | Analysis of sign-up rates and attendance at interviews | Descriptive statistics |
| | Interview with one programme facilitator per case study school (between 1 - 3 depending on whether facilitator runs session in more than 1 school) | Analysis of sign-up rates and attendance at interviews | Descriptive statistics |

## Data analysis

The following section provides a high-level overview of our data analysis plan - we will provide a more detailed overview in a full statistical analysis protocol which will be produced at a later date.

This pilot trial is not primarily designed to estimate effect sizes or evaluate the impact of the intervention in depth, but is instead focussed on assessing if Face It could and should progress to further stages of more rigorous evaluation.

#### Feasibility, acceptability and evaluability analysis

The primary objective of the pilot trial is therefore to establish the feasibility, acceptability, and evaluability of evaluating Face It. This will be done based on framework and descriptive analysis of quantitative and qualitative data, as described in *Table 2*, which will be assessed based on the monitoring criteria discussed in *Section 4* of this protocol.

In addition to the analyses needed to assess our monitoring criteria, we will conduct analysis of programme administrative data to test whether uptake and retention varies by key participant characteristics, and to test correct treatment assignment. Analysis will be pre-specified in the full statistical analysis plan.

We will conduct descriptive analysis of programme administrative and implementation data to inform assessments of trial arrangements and practice model and suitability to proceed with a full evaluation.

#### Effectiveness analysis

In addition to the analysis of the feasibility, acceptability and evaluability of Face It, we will conduct analysis on the outcomes of the pilot study using the following approach, in order to further inform monitoring criteria and our resulting recommendation to YEF.

Our analysis will help us understand if there is sufficient evidence of impact to justify a larger and more robust efficacy trial. Because this is a pilot study with a small sample size, we will have to interpret any statistical results with caution.

We intend to have one primary outcome (the self-reported, post-programme SDQ), and a number of secondary outcomes. These are measured using the following scales:

#### Primary outcome:

SDQ (total difficulties, post-programme self assessment)

Secondary outcomes (all at both post-programme and 3-month follow up:

- SDQ (3-month follow-up self assessment)
- The Self-Report Delinquency Scale

- Problem Behaviour Frequency Scale
- SDQ (parent assessment)
- The Children's Hope Scale
- The Emotional Regulation Questionnaire
- SWEMWBS
- School Attendance
- School Exclusions

We have conducted preliminary assessments of validity and reliability of these scales and judged these to be appropriate for this pilot trial.

All outcome data will be analysed using an intention to treat (ITT) analysis and linear (or logistic where relevant) regressions - high-level equation model below. We will collect pre-intervention outcomes for all students to increase power and adjust for regression to the mean. Our control vector will include gender, ethnicity, FSM status, pre-intervention outcomes, and allocation reason<sup>29</sup>.

$$Y_{i} = \alpha + \beta_{1} * Treatment + \beta_{2} * Control vector + \epsilon_{i}$$

We will conduct subgroup analysis for the 80% of young people showing externalising behaviour to test whether these outcomes vary from the 20% displaying internalising behaviour.

Additionally, we will produce descriptive statistics for individual survey questions that are most relevant to our outcomes (the full statistical analysis plan will clearly define these).

# Risks to study validity

#### **Spillover**

The risk of spillover arises from the potential for students in the intervention group to discuss the programme with students in the control group, thereby providing the control group with some of the learnings from the intervention. However, we have assessed that the risk of spillover is low, given the intense and targeted nature of the intervention. That is, any effects are likely to emerge as a result of participation in the full programme; we do not expect that students discussing the content outside of programme sessions would provide the same benefits. We do not anticipate that an awareness of parts of the programme by those in the control group, or interactions between those in the treatment and the control is likely to impact on the outcomes being assessed.

School staff are not involved in the delivery of this programme, and the likelihood of spillover through staff will be further reduced by ensuring that teachers do not sit in on or observe

<sup>&</sup>lt;sup>29</sup> Defined as whether they fall into the 80% of externalising behaviour or 20% of internalising behaviour

sessions, and by working with new schools who have not experienced the Face It programme before. For example, pupils in the control group of a school which has worked with Khulisa before may experience elements of the intervention if teachers have previously been exposed to programme elements and include them in their lessons and classroom approach.

# Risk that assessment for eligibility will result in control group not receiving service-as-usual (SAU)

We assess that the risk of this is medium. Many teachers and other intervention providers will not be aware that the student has been referred, but there is a risk that some may be aware and adapt their behaviour as a result. We will assess the impact of this by recording what interventions the control and intervention groups received and whether these are different, as well as looking for evidence as to whether this is influenced by the eligibility assessment.

#### **Attrition**

Some degree of young person attrition from the evaluation is to be expected. We will attempt to minimise the impact of this by:

- Providing incentives such as food to all participants when filling out surveys;
- Avoiding unnecessary follow-up by conducting two periods of follow-up (immediately after programme completion and three months after programme completion) rather than three:
- Ensuring that evaluation activities are designed to be low-impact in terms of burden and time;
- Informing schools with sufficient notice about any planned activities with appropriate information about how useful the evidence created by the study will be; and
- Where needed, utilising the relationships that Khulisa has built with LAs to facilitate access and cooperation.

We will monitor rates of attrition and whether there are differences in rates of attrition based on gender, ethnicity, SES (proxied by FSM status) and baseline outcomes.

#### Qualitative research

#### Participatory panel

We propose adopting a participatory approach to the design of our evaluation materials and in understanding our results. To do this, we will conduct a young person participatory panel in one school to inform our evaluation. This will be a school where Khulisa has previously delivered Face It, but where no delivery as part of this evaluation is taking place.

We will involve a small group of up to five young people who have participated in the Face It programme within the last two years to help co-construct elements of our research. Their

experiences and understanding of the programme will inform our decision-making processes and ensure that we appropriately capture participant experiences of the programme. This process will consist of two in-person sessions as follows:

- Session 1: 2-hour session prior to any qualitative data collection to introduce the
  evaluation and the key aims and sense check evaluation materials including, but not
  limited to, interview information sheets and consent forms, and to ask for advice and
  input into improvements.
- **Session 2**: 3-hour session after completion of data collection to help the evaluation team understand and analyse the qualitative data

The young people will be compensated for their time and expertise with shopping vouchers.

As a result of this approach, some of the evaluation tools may change following the first participation panel. We do not anticipate any fundamental changes to the evaluation plan.

#### Qualitative research activities

We will be conducting qualitative research activities within three case study schools. These three schools will be selected from the five participating schools using a convenience sampling approach, depending on schools' availability and willingness to participate. This method will be used to explore and examine experiences and perceptions of the interventions in depth, in three different contexts and using multiple sources of data. We will explore site-specific characteristics and circumstances that influence the implementation of Face It and how this might vary between schools. We will use:

- a) In-person interviews with young people in the intervention group
- b) In-person interviews with parents/caregivers of young people in the intervention group
- c) Online interviews with key school staff who manage the relationship with Khulisa
- d) Online interviews with programme facilitators

#### a) In-person interviews with young people in the intervention group

We will conduct in-person interviews with young people from the intervention group within six weeks after the programme finishes to understand young people's own perceptions and personal experiences of the programme. We will identify 12-18 students (4-6 students per case study school) to participate using a combination of convenience and purposive sampling. As part of the convenience approach we will draw interviewees based on recommendations from the teacher responsible for the relationship with Khulisa and students' availability and willingness to be interviewed. In addition to this, using purposive sampling, we will aim to sample participants across a range of key criteria, namely, gender, school, year group, ethnicity, FSM status, and whether young people display primarily internalising or externalising behaviours. The interviews will either be paired or individual
depending on the feedback that the participatory panel gives and dependent on the young people's own preference.

Interviews will be between 45-minutes and 1-hour in length, will take place at school during the school day, and will be audio-recorded (with consent) and transcribed. Young people will be offered a £10 shopping voucher for compensation for their time and knowledge. Interview guides will be developed in collaboration with Khulisa, and we will seek input from the young person participatory panel (see above) regarding key areas to cover and elements to consider or avoid during interviews. The topic guides for young people will be participant-led to allow the researcher to form a stronger rapport with the participant and generate more in-depth data. This means that topic guides will include a series of prompts relating to the research objectives, rather than representing a predefined list of questions, allowing the researcher to shape the interview based on the participant's responses.

Interview topic guides are likely to focus on the following research questions:

- 1. Acceptability of the programme (Do young people value the programme and feel the content and delivery are appropriate to their needs?)
  - a. What participants' experiences of participating in the programme were
  - b. What participants thought about programme content
  - c. What participants thought about programme delivery
- 2. Programme outcomes (Does Face It show sufficient promise in terms of improvements in key outcomes (resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions) to justify a subsequent efficacy trial?)
  - a. What are the perceived impacts of the programme for young people on resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions?
- 3. Mechanisms (What do young people's perceptions of the programme suggest about possible mediators and moderators?)
  - a. What the perceived mechanisms of change are for young people
  - b. Whether other factors (separate from the programme) contributed to identified changes
- 4. Feasibility: Fidelity of programme (Can Face It recruit and retain sufficient numbers of young people from the target population and deliver the programme with fidelity?)
  - a. What is the degree of young people's engagement with programme activities?

#### b) In-person interviews with parents/caregivers

We will conduct in-person interviews with parents/caregivers of young people in the intervention group in one school around six weeks after the programme finishes to understand the perceived evaluability, acceptability and impact of the intervention. We will use a voluntary response sampling approach - parents/caregivers will be invited to a drop in session, with shopping voucher incentives included as compensation for parents/caregivers' time and knowledge. Evaluation staff will be on hand to conduct up to five interviews with caregivers.

The time frame stated above is indicative - we will be flexible with scheduling the drop in session, aiming to align it with a time where caregivers are already in school (e.g. for parents evenings) to maximise participation. This represents an exploratory part of our approach: this activity will be tested in only one case study school to determine the feasibility of including parent/caregiver views in the larger trial and to understand potential barriers to using this approach. We recognise that there is a risk of a low response rate, and are conducting this activity to assess whether it might be possible in any future trial.

Interviews will be audio-recorded with each participant's permission and then transcribed. Interview topic guides will be developed in collaboration with Khulisa, but are likely to focus on the following research questions:

- 1. Evaluability: Acceptability of data collection (Do we have enough confidence in the feasibility of a randomised controlled trial (RCT), particularly in terms of recruitment into evaluation, randomisation and outcome data collection, to justify a continuation of the efficacy trial past this pilot trial?)
  - a. Are interviews and surveys seen as acceptable?
  - b. How can we optimise qualitative and quantitative data collection from caregivers?
  - c. Why participants chose to participate in interviews
  - d. Why participants think others may choose not to participate
- 2. Acceptability: (Do parents/caregivers find programme delivery acceptable?)
  - a. Is the programme content acceptable to parents/caregivers?
  - b. Is the programme delivery acceptable to parents/caregivers?
  - c. What participants' impressions of YP experience of the programme are
- 3. Programme outcomes: (Does Face It show sufficient promise in terms of improvements in key outcomes (resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions) to justify a subsequent efficacy trial?)
  - a. What are the perceived impacts of the programme on young people's resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions?
  - b. What the perceived mechanisms of change for identified outcomes are

## c) Online interviews with key school staff who manage the relationship with Khulisa

The successful delivery of interventions is often reliant on the engagement of key stakeholders, so it will be important to explore the attitudes of key school staff towards the programme as well as key behaviours and decisions that may have affected programme implementation.

We will interview three members of staff (one from each case study school) around eight weeks after the programme finishes to understand the perceived feasibility, acceptability,

evaluability and impact of the intervention. Interviews will be conducted online, audio-recorded with participants' permission and then transcribed. Interview topic guides will be developed in collaboration with Khulisa, but are likely to focus on the following research questions:

- 1. Feasibility: (Can Face It recruit and retain sufficient numbers of young people from the target population and deliver the programme with fidelity?)
  - a. What school staff perception of the referral process was
  - b. Whether staff were able to identify eligible participants easily
- 2. Acceptability: (Do teachers find programme delivery acceptable?)
  - a. Is programme content and delivery acceptable (e.g. taking children out of lesson time)
  - b. What the facilitators and barriers to effective programme delivery are
- 3. Evaluability: (Do we have enough confidence in the feasibility of a randomised controlled trial (RCT), particularly in terms of recruitment into evaluation, randomisation and outcome data collection, to justify a continuation of the efficacy trial past this pilot trial?)
  - a. Acceptability of randomisation
  - b. What staff members' experiences of participating in the evaluation were
- 4. Programme outcomes: (Does Face It show sufficient promise in terms of improvements in key outcomes (resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions) to justify a subsequent efficacy trial?)
  - a. What are the perceived impacts of the programme on young people's resilience, emotional regulation, social and emotional wellbeing, school attendance and school exclusions?
  - b. Whether they or their colleagues have reported any differences in behaviour among young people

#### d) Online interviews with programme facilitators

We will conduct interviews with 3-6 programme facilitators approximately two weeks after the programme finishes to help us to understand whether the programme was delivered as intended, and to identify any facilitators and barriers to delivery.

Interviews will be conducted online, audio-recorded with participants' permission and then transcribed. Interview topic guides will be developed in collaboration with Khulisa, but are likely to focus on the following research questions:

- 1. Feasibility: Fidelity (Can Face It recruit and retain sufficient numbers of young people from the target population and deliver the programme with fidelity?)
  - a. Can Face It be delivered with fidelity?
  - b. What factors affect fidelity?
  - c. What variations in delivery are appropriate for effective implementation?

- 2. Acceptability: (Do young people value the programme and feel the content and delivery are appropriate to their needs? Do teachers and caregivers find programme delivery acceptable?)
  - a. Is Face It acceptable to young people at risk of youth violence?
  - b. Does participation in a randomised evaluation affect participants' views of the intervention? If so, how?
  - c. Does acceptability vary by ethnicity and race?
  - d. Is the programme acceptable to teachers?
  - e. What factors affect acceptability?
  - f. How could the programme be adapted to increase acceptability?
- 3. Evaluability: (Do we have enough confidence in the feasibility of a randomised controlled trial (RCT), particularly in terms of recruitment into evaluation, randomisation and outcome data collection, to justify a continuation of the efficacy trial past this pilot trial?)
  - a. Is data collection possible and sufficient?
  - b. What factors affect ease of data collection and completeness and quality of data?
  - c. How could the approach to data collection be improved to increase ease, completeness and quality?
  - d. Do practitioners feel that the evaluation impacts on intervention delivery? If so, what elements of the evaluation affect delivery quality?
  - e. Is randomisation acceptable to practitioners & teachers?
  - f. What factors affect acceptability?

#### **Qualitative analysis**

All interview recordings will be transcribed verbatim to ensure accuracy and facilitate subsequent analysis. Transcripts will be anonymised by assigning unique identifiers to each participant, replacing their names or any identifying information.

The research team will immerse themselves in the data before starting the data management and analysis approach. The team will adopt a framework approach to analysis, whereby the key themes emerging from both the research questions and the data are incorporated into an analytical framework where each column represents a subtheme and each row a participant. The interview data is then charted (summarised) into that framework in a comprehensive and systematic way. Once the data management stage is complete, the research team will use the framework to carry out the analysis. This will involve looking at each theme in turn and exploring the range of views held under that theme with a view to developing categories. This will be done by grouping the views into clusters and exploring the properties of each of these clusters until clear categories can be developed. Given the nature of the pilot study and the size and likely diversity of the sample, it is highly likely that the majority of the analysis will be descriptive and aim to clearly map out the range and diversity of views that exist within each participant population on the key areas relevant to the research questions. However, where possible the researchers will proceed to a higher

level of analysis and aim to look for patterns and linkages in the data, as well as explanations.

Verbatim participant quotations and case examples will be used to provide evidence and exemplify the theme(s) discussed.

Quality assurance will be provided by an experienced qualitative researcher.

# 6. Cost evaluation - data collection and reporting

We will report the cost of delivering the intervention in the final report, following YEF costing guidance. We will:

- Use a bottom-up costing approach and break costs down into: prerequisites, set-up costs, and recurring costs.
- We will report the total cost for a typical single cohort receiving the intervention for one round of delivery and the costs per participant for one round of delivery, assuming full compliance. The programme will be delivered within 5 schools, twice within each school, to two different groups of young people (to one group of Year 9s, and to one group of Year 10s). Depending on heterogeneity in costs across cohorts, we will either report average costs, or select a case which we think is most representative of the costs we expect to be incurred in future, typical rounds of delivery.

The organisations and practitioners involved in delivery are Khulisa and the intervention schools. To report cost at the end of this study, we have produced a template for these organisations to complete, covering staff costs, equipment/materials costs, programme procurement costs, and buildings and facilities costs. This template has been reviewed by Khulisa.

We expect most costs to fall within the following two categories:

- Staff cost: cost of practitioners, supervisors, and managers involved in delivering Face It.
- Programme procurement costs: the cost for Khulisa to train and supervise staff, as well as to produce and provide the programme-specific materials required to deliver the programme.

## 7. Planned outputs

The final output of this pilot trial will be a publicly accessible report summarising the evidence for each of the research questions and making a recommendation to YEF about whether to proceed to a full-scale efficacy trial based on a holistic look at the evidence as a whole, highlighting any discrepancies between data sources.

This will involve triangulating information from a range of qualitative and quantitative data sources, from a range of relevant stakeholders comprising young people, parents, school staff, and intervention delivery staff.

## 8. Ethics and data protection

#### **Ethics**

#### Overview

This trial was self-assessed as being high risk due to the inclusion of high risk participants in the form of vulnerable young people. As a result we sought ethical approval from an independent panel of external experts with experience of working with vulnerable children and experience with safeguarding and child protection.

The independent ethics review committee (ERC) reviewed the following information:

- Ethical review form
- Consent forms and information sheets for young people and parents/caregivers of young people
- Student interview topic guide
- Safeguarding and distress protocol

The ERC discussed any issues raised by the research with The Lab with the aim of finding solutions that meet ethical requirements. The reviewers and the project manager agreed solutions to any outstanding issues, and the resulting changes to the way the project is being implemented have been included on the ethics form. The ERC was happy to approve the project with the inclusion of these amendments.

If there are substantial changes while the research or evaluation is being implemented, the ethics form will be revised and the revisions agreed with the ERC.

We conducted a separate internal ethical review for the materials for the participatory panel, as we have judged this to be a separate package of lower risk work. This is because:

- We will be asking young people to comment on our proposed materials and approach rather than on the intervention in detail. This means that any personal reflections and experiences will be limited
- Panel members' views and/or data won't be written up into outputs in the same way
  as material from the evaluation. Instead, they will just shape the evaluation that we
  deliver and the analysis that we conduct.

The participatory panel materials were approved through an internal ethics review process.

#### **Informed Consent**

The Head Teacher or other suitable member of each participating school's Senior Leadership Team will provide written consent for the school to participate in this study. This will take place prior to the Lab/Khulisa receiving any referral data.

We will provide parents/caregivers of young people with an information sheet and withdrawal form, providing the opportunity to withdraw their child from the evaluation prior to seeking consent from young people. Any parents/caregivers who don't want their child's data to be used in the evaluation will be able to withdraw their child from the trial prior to any data collection. No data will be gathered on the child and the child will not participate in the Face It programme.

We will obtain written consent from young people to take part in the evaluation prior to baseline data collection. We will then also obtain written consent at every data collection activity (embedded within surveys, at the beginning of YP interviews, at the beginning of all other stakeholder interviews - parents/caregivers, facilitators, key school contact). The only exception to this will be in special circumstances (e.g. where participants have accessibility needs, such as severe dyslexia); in these instances we will seek verbal recorded consent.

We will take steps to ensure consent is fully informed, including comprehensive, but accessible, information sheets, going over the information sheet content verbally, and giving plenty of opportunity for participants to ask any clarifying questions. The information sheets will include information about the nature and purpose of the study, the organisations involved, what data will be collected, what will happen to it and why, and offer participants the opportunity to opt out of the research. The information sheets will be sent via email and will include a link to the privacy notice and will explain that we will ensure confidentiality and anonymity in reports, providing all information in clear, accessible language. Where we think consent is not being made on an informed basis we will not continue with data collection activities for that participant.

We will review the information sheets and consent forms with the young person participatory panel to ensure that the information is clear and accessible.

At any point until 1st May 2024, participants or their caregivers can withdraw their or their child's participation from the trial. If participants withdraw from the trial before any of their personal data is shared with the Lab, then the young person will not participate in the evaluation and no personal data will be shared.

Should we be informed that participants would like to withdraw from the trial after some personal data has been collected we will not collect any additional personal data and will, where possible, delete all of the participant's personal data collected up to that point (other than interview responses that have already been analysed and anonymised).

We will make it clear to participants that we will use their information to inform the findings of our evaluation, which will be incorporated into a report, or other publicly publishable materials. However, no identifying information will be disclosed in any such materials.

#### Safeguarding

Given the potential vulnerability of the young people involved in this evaluation, we have ensured that we have a stringent safeguarding plan in place throughout.

All researchers with any contact with children will have an enhanced DBS check, will have completed NSPCC Safeguarding training, and will familiarise themselves with the BIT Group Safeguarding Policy and the project safeguarding and distress protocol.

Researchers conducting in-person data collection in schools will comply with all school requirements for visitors.

## **Data protection**

We will follow appropriate data protection processes in accordance with BIT processes, including completing a Data Protection and Security Checklist and Data Protection Impact Assessment which have both been reviewed and approved by BIT's legal team.

The legal basis for processing personal data will be legitimate interest and the legal basis for processing special category data will be scientific interest. Article 6(1)(f) of UK GDPR states that "processing is necessary for the purposes of the legitimate interests pursued by the controller or by a third party except where such interests are overridden by the interests or fundamental rights and freedoms of the data subject which require protection of personal data, in particular where the data subject is a child."

The Lab has determined that there is a genuine purpose to process this data. The purpose of processing personal data is to assess whether it will be possible to conduct a full-scale randomised controlled trial evaluation of the Face It intervention, through assessing feasibility, acceptance, and evaluability of the intervention, and estimating initial outcomes of

the intervention. Answering this question will help us, YEF, and the wider education and youth violence prevention sector to better understand effective support to vulnerable young people at risk of exclusion and becoming involved in violence. This will inform the evidence around what works to improve the health, behaviours and life outcomes of young people, particularly those at risk of, or who have engaged in, violent behaviours. Data processing is necessary to complete a robust evaluation. The Lab does not consider that collecting and gathering data for this trial will interfere with individuals' interests, rights or freedoms. The data subjects will include: at-risk youth, caregivers of at-risk youth, the delivery team at Khulisa, and school staff responsible for the relationship with Khulisa.

All data shared with BIT will be processed in line with its data protection policy. A summary of this policy can be found in Annex G. In the analysis, BIT will promote data quality and security through the following measures.

- All variables will be clearly named, coded and labelled before analysis.
- Checks on the data received will be carried out for valid values, range, and consistency against already held data.
- Any modifications to datasets will be recorded in the analysis code, which will be well-annotated.
- Original raw datasets will never be amended.
- Access to the project data will be restricted to project personnel.
- All data stored by BIT will be backed up.

A project privacy notice for this project will be shared with participants and published on the Lab's website.

## Data management

All quantitative and qualitative data will be stored in a secure Google Folder where access is restricted to only researchers conducting the analysis. Data will be deleted upon completion of the project in March 2025.

After the project has been completed, data will be shared with YEF, pseudonymised, and stored in the YEF Evaluation Data Archive. All projects funded by YEF store data in this way. Data in the archives is separated from any identifiable information.

Approved researchers may apply to access YEF data via the Office of National Statistics (ONS) secure research service. This will be accessed via their own project space created in the ONS secure research environment by the ONS. They may apply to the Department of Education and Ministry of Justice to access the linked National Pupil Database-National Police Computer data, and if successful it will be made available here to combine with the YEF evaluation data, using pupil matching reference numbers. Researchers will only be able to access pseudonymised data. All results will be published in a de-identified form.

This enables YEF to assess the impact of their projects long-term, as well as to conduct quality assurance, reanalysis and methodological exploration across the outputs and results

published in the YEF funded evaluation reports; and pooled analysis of data from multiple interventions, to explore what works in different geographic areas and for particular subgroups (e.g. gender, ethnicity, child who have experienced periods of care etc) that may be identified from the data collected from the projects themselves or from the linked administrative datasets.

Further information about this process can be found on the YEF website.<sup>30</sup>

#### Quantitative data

#### Survey data

We will use SmartSurvey to collect the survey data. SmartSurvey produces a spreadsheet where one row is a survey response. This will be used to code the survey outcomes using the methods outlined in the outcome measures table.

Surveys will ask participants to record their name. This enables us to link survey responses with demographic data and other outcome measures. Once survey responses have been linked, participants' names will be removed.

#### ImpactEd and programme administrative data

Khulisa is responsible for providing us with both the ImpactEd and programme administrative data. All data shared with the lab by Khulisa will be received via a secure transfer link (Virtru or Quatrix).

**ImpactEd data** will be collected via ImpactEd, shared with Khulisa who will in turn share it with us. They have used ImpactEd before in the past and are confident the data will be of high quality.

**Programme administrative data** includes the *referral data* and the *programme delivery data* (e.g. attendance sheets, fidelity checklists). *Referral data* will be collected via an online form (located on FormAssembly) completed by school staff. Khulisa will download the data in a spreadsheet and share the relevant data with the lab. *Programme delivery data* will be collected via Khulisa, and shared with the lab.

#### **Qualitative data**

#### Interview transcripts

Interview recordings will be uploaded to McGowan for transcription. All interview recordings will be transcribed verbatim to ensure accuracy and facilitate subsequent analysis.

<sup>&</sup>lt;sup>30</sup>https://youthendowmentfund.org.uk/wp-content/uploads/2021/07/YEF-Data-Guidance-Projects-and-Evaluators.pdf

Transcripts will be anonymised by assigning unique identifiers to each participant, replacing their names or any identifying information. Transcripts, observation notes, and any additional relevant documents will be securely stored in a password-protected file area. Access to the data will be restricted to only project team members involved in the analysis. Recordings will be deleted after completion of the project, in March 2025.

## 9. Racial diversity and inclusion

The Lab is committed to conducting research in which equality, diversity and inclusion principles are firmly embedded across all stages of this evaluation, including the design, recruitment, data collection, and analysis.

i) Groups included in the programme and evaluation. Prior to eliciting student referrals from schools, Khulisa will conduct work against unconscious bias with relevant staff members using material developed with UNLRN. This will consist of educating staff about unconscious bias and sharing strategies to minimise this when considering which students to refer to the programme. Khulisa will also work to refine their target population and materials communicating this to schools to ensure that the most appropriate young people are referred to the programme.

We will work with Khulisa to develop a final sampling frame that meets the primary needs for our evaluation. For example, our primary sampling criteria for interviews will be young people who have engaged with Face It, and we will purposively sample young people across the following key characteristics (as far as is possible within our sample size): ethnicity, gender (including non-binary descriptors), year group, school, free school meal status (as a proxy for socio-economic status), and whether young people display primarily internalising or externalising behaviours.

#### ii) Inclusivity during the design of the evaluation

We propose adopting a participatory approach to the design of our evaluation materials and in understanding our results. By including a small group of young people (up to five) who have previously participated in the Face It programme within the last two years, we will protect against researcher bias in the design of elements of our research. Their experiences and understanding of the programme will inform our decision-making processes and ensure that we appropriately capture participant experiences of the programme.

These young people will be selected using convenience sampling, but, if possible, we will aim for the group to represent a range of demographic characteristics.

iii) Inclusivity during recruitment. The Lab will ensure that inclusive practices are central to our *recruitment process* and that participant wellbeing is promoted by (i) being considerate of the sensitivity of the topic area during recruitment - e.g. providing the option of a paired or individual interview, within a school setting or online (ii) providing young people with welcoming and accessible information sheets, co-designed with young people on your participatory panel, that gives all of the information about data security, anonymity and the reasons for undertaking research (iii) ensuring that information is accessible to young people who struggle to engage with written text, such as through offering a hard copy version of any documentation with a yellow overlay for individuals with severe dyslexia, or providing an audio recording of information sheets and other relevant documentation (iv) we will offer flexible interview times that allow for different groups and individuals the opportunity to participate (see next section).

#### iv) Inclusivity during data collection

For the delivery of Face It, Khulisa works to ensure racial diversity of practitioners in a manner that is representative of the demographics of the target school. For the evaluation, we will:

- Minimise power imbalance: Negative effects of power-imbalance can lead to false, distorted or limited information being disclosed, or the interviewee relating what they think the interview wants to hear. To protect against this BIT will: (i) collect data through individual or paired interviews; (ii) include tools within our enquiry process that ensure that people participate in a more equitable way that is not simply through verbal response. Researchers will endeavour to ensure inclusive facilitation through displaying empathy and respect for participants' views and experiences.
- 2. Mitigate access issues: Enabling inclusive access to interviews requires considering the factors that limit attendance. Access issues could include a lack of time during the day to attend sessions, or distance from an in-person session. The Lab aims to enable wide access to the sessions by offering to conduct interviews within a school setting wherever possible. We could also offer remote sessions if young people prefer, making accessing the session easier. The use of Google Meets does not require new software to be installed and participants can join Google Meets meetings through telephone connection, so do not need internet access. We will offer to use other software such as Microsoft Teams or Zoom if this is more accessible to the individual.
- 3. **Training for researchers:** Prior to conducting interviews, researchers will complete the NSPCC's Introduction to safeguarding and child protection training and complete a pre-interview workshop on interviewing best-practice with NJ Research Ltd.

**iii) Wellbeing and safety during interviews**. The Lab is conscious that young people who engage in the evaluation could be vulnerable to negative and stressful impacts of the research process. The Lab will work to ensure the wellbeing and psychological safety of individuals during data collection by:

- 1. Designing interview questions to minimise harm and maximise comfort: The Lab will maximise wellbeing and minimise harm during qualitative data collection by (i) structuring topic guides to begin the interview with simpler questions which can build in complexity and difficulty as the participant becomes more comfortable and rapport develops, (ii) depersonalising questions to elicit comfort and stronger answers (e.g. instead of 'what do you hate about X', ask 'lf you had a magic wand, what 3 things would you change about X to make it easier?'), (iii) being aware of tension, discomfort or distress during the interview, repeating that the interview can be stopped if participants wish, and repeatedly asking participants if they want to continue, (iv) ensuring that researchers are aware of places to signpost participants and offering this information, and (v) auditing the questions for their sensitivity within the context before the interview.
- 2. Allowing the participants to choose their environment for participating: Where possible, the Lab will allow the interviewees to make decisions about the interview setting at their home, a public place or over the phone, enabled by the online conference format.
- 3. Reminding participants of anonymity and data security: The Lab will endeavour to minimise stress by reminding participants that data collection is fully anonymous and all identifiable information will be removed from the transcripts and report. It often helps to say what this means, e.g. 'We will describe you as a year 9 student from a school in London'. The Lab can also offer the chance for them to check over the anonymised transcript.
- 4. Incorporating the views of the participatory panel: The Lab will seek the views of the participatory panel on elements relating to interview logistics, such as whether to proceed with individual or paired interviews, in order to ensure that arrangements are acceptable to young people.

**Inclusivity during data analysis:** The Lab feels it is also important to preserve EDI principles within the data analysis stage too. This will be achieved by engaging the participatory panel to cross check our analysis and emerging themes, to ensure that we have an inclusive and informed approach to analysis.

## 10. Risks

We have identified the following risks.

| Risk | Impact | Likelihood | Mitigation |
|---|---|---|---|
| Exclusion outcome confounded with intervention (i.e. if schools are less likely to exclude pupils while they are on the programme) | Medium | Low | Unlikely as schools have previously excluded pupils receiving Face it, and many teachers will not be aware of the programme. |
| Spillover between treatment and control participants | Medium | Low | Ensuring that teachers do not sit in and observe programme sessions will reduce the chance of spillover. Working with new schools who have not experienced the Face It programme before, where teachers will not be familiar with the programme content will also reduce the likelihood of spillover. For example, pupils in the control group of a school which has worked with Khulisa before may experience elements of the intervention if teachers have previously been exposed to programme elements and include them in their lessons and classroom approach. |
| Unconscious bias in pupil referrals (i.e. disproportionately referring children of minority ethnic backgrounds based on unconscious bias | Medium | Medium | There is potential for unconscious bias due to the use of teacher referrals. However, we will aim to minimise the likelihood of this by using a detailed referral form developed and used by Khulisa. The form prompts referrals to consider multiple factors such as students' current needs and adverse childhood experiences, reducing the likelihood of referral solely due to bias. In addition, prior to referrals, Khulisa will provide schools with resources developed with charity partner Chasing Prospects and consultants UNLRN which aim to tackle unconscious bias. As part of the pilot evaluation, we will monitor this risk by monitoring the characteristics of young people being referred to the programme, and discuss this concern with practitioners as part of qualitative interviews. |

| Non-compliance by staff with random assignment | High | Medium | We will ensure that school and delivery partners are aware of the implications of non-compliance with randomisation prior to recruitment. We will conduct randomisation close to the start of delivery, by conducting randomisation separately for each school. We will also issue schools with an information sheet reiterating the importance of compliance. We will also encourage Khulisa to communicate the importance of compliance with randomisation in discussions with schools. |
|---|---|---|---|
| Low recruitment and retention of schools | Medium | Medium | School recruitment and retention will be a responsibility of Khulisa. Khulisa will aim to reduce this risk by initiating discussions early with schools and working to maintain positive relationships with schools. |
| Low recruitment of eligible young people within schools | Medium | Low | Face It is typically oversubscribed and there are processes in place to monitor the trajectory of recruitment and retention |
| High dropout rate from evaluation among young people | Medium | Medium | Provision of incentives for survey completion sessions for both the intervention and control groups. |
| Sites (or participants within sites) will not engage with evaluation activities | Medium | Medium | Some amount of attrition is to be expected in all evaluations. We have several strategies that aim to minimise attrition, which include: • ensuring buy-in from the Headteacher and/or senior leadership team; • identifying a specific individual responsible for the relationship between the school and Khulisa, and for communications with the Lab; • ensuring that evaluation activities are designed to be low-impact in terms of burden or time, by avoiding unnecessary data collection, and incentivising activities where appropriate; • informing sites with sufficient notice about any planned activities with appropriate information about how useful the evidence created by the study will be; and • where needed, utilising the relationships that Khulisa has built with LAs and schools to facilitate access/cooperation. |

## 11. Timeline

This pilot study is expected to last 18 months from April 2023 to September 2024, subject to appropriate school recruitment and young person referral. While the Lab will endeavour to facilitate this, these processes are ultimately out of our direct control.

| Phase | Activity | Description of activities during phase | Led by | Target date |
|---|---|---|---|---|
| Project set up | Delivery<br>Planning | Internal delivery plans and project management tools developed | Khulisa | July 2023 |
| Froject set up | | Recruitment and training completed | Khulisa | Aug 2023 |
| | Evaluation design | Protocol published and detailed internal plans and project management tools development | The Lab | July 2023 |
| | | Development of surveys, interview guides and other data collection tools | The Lab | July 2023 |
| | | Statistical Analysis Plan developed | The Lab | Sep 2023 |
| | School recruitment | Development of materials for recruitment of schools explaining evaluation, randomisation etc. | Khulisa | April 2023 |
| | | Target number of schools agreed to participate in the evaluation | Khulisa | By July 2023 |
| | Participatory panel | Participatory panel session 1 | The Lab | September 2023 |
| | Young<br>person<br>recruitment | At least 160 eligible young people referred to the programme | Khulisa | Oct 2023 |
| | | At least 160 young people randomised into intervention or control | Joint | Nov 2023 |
| Project<br>delivery and<br>data collection | Baseline<br>data | Young person baseline survey for cohort 1 (Autumn term) | The Lab | Sep 2023 |
| | collection | Young person baseline survey for cohort 2 (Spring term) | The Lab | Jan 2024 |
| | | Parent/caregiver baseline survey for | The Lab | Sep 2023 |

| cohort 1 Parent/caregiver baseline survey for cohort 2 Baseline attendance and exclusion data Delivery Delivery for schools in cohort 1 Programme data on retention, fidelity etc. for cohort 1 Programme data on retention fidelity etc. for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in choort 3 Interviews with you | | | | | |
|---|---|---|---|---|---|
| cohort 2 Baseline attendance and exclusion data Delivery Delivery for schools in cohort 1 Khulisa Oct 2023 Delivery for schools in cohort 2 Khulisa Feb 2024 Programme data on retention, fidelity etc. for cohort 1 Interviews with young people in cohort 1 Programme data on retention fidelity etc for cohort 1 Interviews with young people in cohort 2 Young people end-of-programme survey for cohort 2 Young people end-of-programme asurvey for cohort 2 Young people end-of-programme survey for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in cohort 2 Interviews with young people in The Lab Mar 2024 Interviews with young people in Cohort 2 Interviews with young people in The Lab March 2024 cohort 1 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey The Lab March 2024 cohort 1 Young person follow-up survey The Lab May 2024 cohort 1 Young person follow-up survey The Lab May 2024 cohort 2 Parent/caregiver follow-up survey The Lab May 2024 cohort 2 Attendance and exclusion data cohort 3 Analysis of quantitative write up Produce descriptive statistics of adding data collection | | | cohort 1 | | |
| Delivery Delivery for schools in cohort 1 Khulisa Oct 2023 Delivery for schools in cohort 2 Khulisa Feb 2024 Post-intervention data collection Programme data on retention, fidelity etc. for cohort 1 Interviews with young people in Cohort 1 Programme data on retention fidelity etc for cohort 1 Programme data on retention fidelity etc for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in Cohort 2 Interviews with young people in Cohort 2 Interviews with young people in Cohort 2 Interviews with young people in Cohort 2 Interviews with young people in Cohort 1 Programme data on retention fidelity etc for cohort 2 Interviews with young people in Cohort 2 Interviews with young people in The Lab Mar 2024 Cohort 1 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey The Lab March 2024 Cohort 1 Young person follow-up survey The Lab May 2024 Cohort 2 Parent/caregiver follow-up survey The Lab May 2024 Cohort 2 Parent/caregiver follow-up survey The Lab May 2024 Cohort 2 Attendance and exclusion data Chulisa Chulisa Cohort 2 Attendance and exclusion data Chulisa Chulisa Cohort 2 Attendance and exclusion data Chulisa Collection | | | | The Lab | Jan 2024 |
| Delivery for schools in cohort 2 Khulisa Feb 2024 Post-interve ntion data collection Programme data on retention, fidelity tet. for cohort 1 Young people end-of-programme survey for cohort 1 Interviews with young people in cohort 1 Programme data on retention fidelity etc for cohort 1 Programme data on retention fidelity etc for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in The Lab Mar 2024 Cohort 1 Parent/caregiver follow-up survey The Lab March 2024 Cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey The Lab May 2024 Cohort 2 Parent/caregiver follow-up survey The Lab May 2024 Cohort 2 Parent/caregiver follow-up survey The Lab May 2024 Cohort 2 Attendance and exclusion data Khulisa May 2024 Cohort 2 Attendance and exclusion data Cohort 2 Produce descriptive statistics of and report write up Produce descriptive statistics of admin data collection | | | | Khulisa | Dec 2023 |
| Post-interve ntion data collection Programme data on retention, fidelity etc. for cohort 1 Young people end-of-programme survey for cohort 1 Interviews with young people in cohort 1 Programme data on retention fidelity etc for cohort 2 Young people end-of-programme survey for cohort 2 Young people end-of-programme survey for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in chall shall | | Delivery | Delivery for schools in cohort 1 | Khulisa | Oct 2023 |
| ntion data collection Young people end-of-programme survey for cohort 1 | | | Delivery for schools in cohort 2 | Khulisa | Feb 2024 |
| survey for cohort 1 Interviews with young people in cohort 1 Programme data on retention fidelity etc for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in cohort 2 Interviews with young people | | ntion data | | Khulisa | Dec 2023 |
| cohort 1 Programme data on retention fidelity etc for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in cohort 2 The Lab March 2024 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 The Lab May 2024 Attendance and exclusion data cohort 2 The Lab May 2024 Attendance and exclusion data cohort 2 The Lab data cohort 2 | | | | The Lab | Dec 2023 |
| etc for cohort 2 Young people end-of-programme survey for cohort 2 Interviews with young people in cohort 2 Interviews with young people in cohort 2 3 month follow up Young person follow-up survey cohort 1 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 The Lab May 2024 May 2024 The Lab May 2024 | | | | The Lab | Jan 2024 |
| Survey for cohort 2 Interviews with young people in cohort 2 Interviews with young people in cohort 2 Interviews with young people in cohort 2 The Lab March 2024 Young person follow-up survey cohort 1 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 Analysis of quantitative data Produce descriptive statistics of admin data The Lab May 2024 Khulisa May 2024 The Lab May 2024 | | | | Khulisa | Feb 2024 |
| cohort 2 3 month follow up Parent/caregiver follow-up survey cohort 1 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 The Lab May 2024 May 2024 Experiment of the Lab May 2024 The Lab Chulisa May 2024 | | | | The Lab | Feb 2024 |
| follow up Parent/caregiver follow-up survey cohort 1 Parent/caregiver follow-up survey cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 The Lab May 2024 Parent/caregiver follow-up survey cohort 2 The Lab May 2024 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 The Lab May 2024 Data analysis and report write up Analysis of quantitative data The Lab and another final data collection The Lab another final data The Lab another final data The Lab another final data The Lab another final data | | | | The Lab | Mar 2024 |
| Cohort 1 Attendance and exclusion data cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 Attendance and exclusion data cohort 2 Data analysis and report write up Analysis of quantitative data Cohort 1 Khulisa May 2024 Khulisa May 2024 The Lab 3 months after final data collection | | | | The Lab | March 2024 |
| Cohort 1 Young person follow-up survey cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 Cohort 2 Analysis of and report write up Analysis of data Cohort 2 Produce descriptive statistics of admin data The Lab May 2024 Khulisa May 2024 The Lab Cohort 2 The Lab T | | | | The Lab | March 2024 |
| Cohort 2 Parent/caregiver follow-up survey cohort 2 Attendance and exclusion data cohort 2 May 2024 Khulisa May 2024 Cohort 2 Data analysis and report write up Analysis of quantitative data Produce descriptive statistics of admin data The Lab 3 months after final data collection | | | | Khulisa | March 2024 |
| Cohort 2 Attendance and exclusion data cohort 2 May 2024 Cohort 2 Data analysis and report and report write up Analysis of quantitative data Cohort 2 The Lab 3 months after final data collection | | | | The Lab | May 2024 |
| Data analysis Analysis of quantitative write up Cohort 2 Produce descriptive statistics of admin data The Lab 3 months after final data collection | | | . , | The Lab | May 2024 |
| and report quantitative admin data final data write up data final data collection | | | | Khulisa | May 2024 |
| Apply Statistical Analysis Protocol to The Lab 3 months after | and report | quantitative | | The Lab | final data |
| | | | Apply Statistical Analysis Protocol to | The Lab | 3 months after |

| | outcomes data | | final data collection |
|---|---|---|---|
| | Internal and external quality assurance | The Lab | 4 months after final data collection |
| Analysis of qualitative data | Analysis of transcripts from interviews with young people | The Lab | 3 months after final data collection |
| | Analysis of transcripts from interviews with parents/caregivers | The Lab | 3 months after final data collection |
| | Analysis of transcripts of interviews with practitioners and pastoral leads | The Lab | 3 months after final data collection |
| Participatory panel | Participatory panel session 2 | The Lab | Following initial analysis, prior to reporting |
| Quantitative<br>and<br>qualitative<br>analysis | Quality assurance | The Lab | 4 months after final data collection |
| Drafting and publication | Draft report submitted for external quality assurance | The Lab | 6 weeks after<br>completion of<br>QA of analysis |
| | Quality assurance | The Lab | 2 weeks after above |
| | Final revisions and publication | The Lab | 1 month after above |

#### Annexes

## Annex A: Summary of Face It programme using the TIDieR framework

Name: Provide a name or Face It phrase that describes the intervention. Why: Describe any Due to the high levels of trauma typically experienced by rationale, theory, or goal of Khulisa's participants, Face It is scaffolded around the elements essential to the trauma-informed methodologies like Bruce Perry's intervention. neurosequential model (Perry 2006, 2009). According to this model, in order to manage the impact of trauma in the brain, participants first need help to 'regulate' their emotions, to calm and ground them sufficiently to reduce their level of arousal (amygdala hijack). This then enables them to 'relate' in a way that enables them to trust others to keep them safe to try new things. Only then is it possible to 'reason' with them, to work with the cognitive part of the brain. The process of how change happens set out by Bruce Perry's model also ties into our Theory of Change. Khulisa's theory of change supports the importance of six clusters of social and emotional skills outlined in the EEF's Spectrum Framework to support young people's social and emotional wellbeing and positive longer-term life outcomes (Education Endowment Foundation, 2017). These competencies are inter-connected and at times overlapping. The aim of Khulisa's programme is to develop this broad spectrum of social and emotional skills, but improved resilience, coping skills, and self regulation are prioritised as key short-term outcomes as in order to improve social and emotional wellbeing, we must first improve young people's coping skills, emotional regulation and resilience. Heading straight for the 'Reasoning' part of the brain is unlikely to be successful if the young person is dysregulated,

stressed and disconnected. First, the person needs help to regulate and calm their flight / fight / freeze responses and build resilience and coping skills to lay the foundation for them to engage with more challenging parts of the programme and

wider life, in order to improve levels of wellbeing.

What - Materials: Describe any physical or informational materials used in the intervention, including those provided to participants or used in intervention delivery or in training of intervention providers. Provide information on where the materials can be accessed.

Before they ever deliver a programme, facilitators are given access to:

- 1. The full programme methodology
- 2. The scaffolding process
- An example high level lesson plan that gives a skeleton overview of the process and content of a programme, to enable them to gradually immerse themselves in the detail that sits behind it.
- 4. A recommended reading list on each of the theoretical concepts that underpin the programme.

In the set up phase of the programme, they have access to the following documents:

- Our participant profile- shared with schools to support the referral process.
- A draft letter to parents sent out by schools.
- A safer recruitment doc that explores our initial safeguarding processes and procedures with Partners
- A Programme Venue Health and Safety Risk Assessment

Supporting materials for the delivery of the programme:

- Lesson plan templates these are edited for each programme.
- A programme fidelity checklist highlighting the core elements every Face It programme should have
- A list of icebreakers and games.
- The poems and games we use on the programme.
- 1 page guides to key activities.
- Handouts to share with participants as part of the programme activities.

#### What - Procedures:

Describe each of the procedures, activities, and/or processes used in the intervention, including any enabling or support activities.

**Pre-programme one-to-one session:** Discussion of pre-programme survey

**Pre-programme group session**: The focus of this session is around building a sense of safety. The activities are based on creating rituals and clear boundaries. By the end of the session: YP understand how to check in authentically so we can respond to their needs, YP empowered to do/not do the programme.

#### 5-day intensive programme:

- Day 1
  - Intro and contracting: Participants feel involved, will have contributed to the group code, & be contained by the knowledge that this is their space.
  - Understanding me: Participants start identifying

- their habits and understand that the journey to change can be challenging, identify the impact of beliefs on our behaviour, understand others' perspectives & experience.
- Introduction to triggers: Participants understand that when we are triggered it can affect how we perceive things around us as well as our reactions

#### Day 2

- Triggers continued: Participants understand the power of triggers and the effects acting on them can have and develop some negotiation skills.
- Emotional literacy: Participants will understand their physiological and emotional responses when triggered, have a better understanding of their own and others' experiences of dysregulation, understand the relationship between emotional responses & brain development, setting the scene for coping strategies.
- Embedding emotional literacy: Participants will be able to differentiate between observable behaviours and the underlying emotions or triggers, develop their ability to empathise and communicate effectively by considering the underlying emotions in themselves & others. They will also practise self-awareness.

#### Day 3

- Exploring challenges: Participants understand different types of violence, and the distinctions between them. They will explore less apparent types of violence and begin to recognise the common thread of power & control that links different types of violent behaviour.
- Challenges continued: Participants will apply their understanding of different types of violence to real-life scenarios, practice empathy by playing different roles in freeze frames and reflect on their own behaviours and attitudes to inferiority/superiority and develop an awareness of how their behaviour can impact their relationships/contribute to conflict.
- Challenge cycle: Participants will realise there is a pattern to violence (it doesn't just happen), start to identify their own pattern of behaviour, recognise they are not alone in their thoughts, feelings, actions and needs and understand

how unmet needs contribute to reactions - all setting the scene for coping skills on day 4.

#### Day 4

- Understanding impact of behaviour & developing coping skills: Participants will gain a deeper understanding of the Challenge Cycle and its impact on others. They will also practice and embed effective strategies to manage challenging situations and emotions building their toolbox of healthy coping mechanisms.
- Accepting my mask: Participants will explore the concept of masks, connect with their challenged selves, express themselves artistically, and engage in meaningful dialogue within a therapeutic and supportive setting.
- Accept and appreciate me: Participants connect with their authentic self, recognise their skills, assets and attributes and consider what's important to them to start the healing process.

#### Day 5

- Asset building: Participants will build their self-esteem, self-worth and their capacity to present positively to others.
- Future focus: Participants will connect with their aspirations, develop a clearer understanding of their past and future, enhance their communication skills, and gain insights into personal growth and decision-making.
- Appreciation and close: Participants will further their self-acceptance, develop their resilience and connect their progress to the overarching learning outcomes, exercise choice and agency, and conclude the day with a sense of reflection and fulfilment.

**Post-programme group session:** The focus of this session is reflection and helping participants to recognise their personal strengths. Appreciation, gratitude and reflective practice enable participants to realise their progress and to consider how they can apply what they've learnt in their daily lives

**Post-programme one-to-one session:** Most significant change discussion, discussion of post-programme survey

**Who:** For each category of intervention provider (such as psychologist, nursing

Khulisa ensures that all facilitators are therapeutically trained in art or dramatherapy so that they have the skills and training required to create 'safe containment' for the group and to assistant), describe their expertise, background, and any specific training given.

continually assess the pace and content of programmes based on participants' needs. There is no minimum level of therapeutic training, but each programme has someone who is therapeutically trained.

All programme managers and associate facilitators receive a stringent 3-day training programme to ensure that they are well-versed in programme content and methodology before they ever deliver a programme. They will also complete levels 2 and 3 safeguarding training. Each programme manager observes and supports 8 programmes as a co-facilitator before they lead a programme of their own.

All facilitators are given access to our written methodology and scaffolding process along with a programme manual setting out key activities corresponding to specific parts of the neurosequential model.

Facilitators receive ongoing support via monthly clinical supervision, fortnightly/monthly supervision with their line manager, monthly group supervision and peer to peer training support every 6 weeks (during half-terms as there will be no delivery). In addition during half-terms/summer provision, Face It offers a weekly optional online session for staff to practise activities together.

Facilitator backgrounds include counselling and youth work, drama and movement therapy, education, education psychology, and dance movement therapy.

How: Describe the modes of delivery (such as face to face or by some other mechanism such as internet or telephone) of the intervention and whether it was provided individually or in a group.

**Pre-programme one-to-one session:** One 60 minute in-person session

**Pre-programme group session:** One 2.5 hour in-person session

**5-day intensive programme**: One intensive 5-day programme delivered in person each day from 9:30-15:30, Monday-Friday

**Post-programme group session:** One 2.5 hour in-person session

**Post-programme one-to-one session:** One 60 minute in-person session

Where: Describe the type(s) of location(s) where the intervention occurred, including any necessary infrastructure or relevant features.

School-based

Khulisa shares a list of programme venue room requirements with schools as part of our service level agreements.

#### When and how much:

Describe the number of times the intervention was delivered and over what period of time including the number of sessions, their schedule, and their duration, intensity, or dose.

The following intervention components are spread over a period of approximately 6 weeks. This estimates one session a week, with a break for half term.

**Pre-programme one-to-one session:** One 60 minute session

**Pre-programme group session:** 2.5 hours **5-day intensive programme**: One intensive 5-day programme delivered each day from 9:30-15:30 Monday-Friday

Post-programme group session: 2.5 hours

Post-programme one-to-one session: One 60 minute

session

**Tailoring:** If the intervention was planned to be personalised, titrated or adapted, then describe what, why, when and how.

Modification within programme description based on ongoing facilitator assessment of group dynamics. For example, facilitators choose an initial icebreaker from a predefined list of options, depending on the dynamic of the group and whether they aim to calm or energise participants.

**Modification:** If the intervention was modified during the course of the study, describe the changes (what, why, when, and how).

To be assessed as part of the pilot trial.

How well (planned): If adherence or fidelity was assessed, describe how and by whom, and if any strategies were used to maintain or improve fidelity, describe them. Our programme delivery is often emergent, and dependent on the emotional regulation and capacity of Khulisa's participants. Throughout each day of the programme various icebreakers, games and energisers are used to assist in the regulation of emotions. This ensures Khulisa's Facilitators can safely contain participants, whilst still providing an opportunity for learning and education.

Our programme balances the flexibility afforded by this emergent process with a very robust methodology and scaffolding process based on Bruce Perry's **neurosequential model** (Perry 2006, 2009). To further ensure programme fidelity and to quality assure our programmes we have identified and closely monitor core milestones and activities every Face It programme should contain. This means that as different as the configuration of programme activities in response to specific needs of the group might be, we will have visibility of and an ability to ensure every Face It programme touches on key milestones that we have identified are central to effecting change. These are reviewed every six weeks as a measure of accountability and quality assurance for the team.

How well (actual): If actual adherence or fidelity was assessed, describe the extent to which the intervention was delivered as planned.

To be assessed as part of the pilot trial.

## Annex B: Khulisa's Theory of Change narrative and diagram

Khulisa delivers intensive social and emotional skills development programmes for young people in schools, pupil referral units, prisons and communities. Programmes are delivered for up to 12 participants at a time over a 6-8 week period. We aspire to only work in organisations where we can deliver training and support for professionals alongside direct delivery. This promotes culture change and an organisation-wide focus on developing and sustaining social and emotional wellbeing. We believe that schools and prisons have a crucial role to play in promoting wellbeing in everything they do, for both young people and the staff who support them.

When we use the term 'social and emotional wellbeing', we mean "the strength and capacity of our minds to grow and develop, to be able to overcome difficulties and challenges and to make the most of our abilities and opportunities" (Young Minds, 2006).

Why focus on Social and Emotional Learning and Wellbeing? Research and evidence clearly shows that social and emotional learning (SEL) and wellbeing is central to successful life outcomes for all young people (Moffitt et al., 2011; Sacker et al., 2007; Gutman et al., 2012; Department for Education, 2011). There is international evidence that SEL reduces mental health issues, prevents criminal behaviour and promotes not only academic achievement, but lifelong learning, satisfaction and success (Cefai et al., 2018; PHE, 2017; WHO, 2012). Evidence shows that SEL is successful for young people from across ethnic, cultural and economic backgrounds and is especially effective for young people from disadvantaged backgrounds (Ceefai et al., 2018; Clarke et al, 2015). The positive impacts of quality SEL are proven to persist over time and deliver strong financial returns on investment (Cefai et al., 2018), with Public Health England reporting a cost benefit ratio of 5:1 (PHE, 2017).

The Context: Despite this evidence, there is inconsistent delivery of SEL in schools, prisons and in the community. We are facing a wellbeing crisis in the UK, with young people reporting the lowest levels of wellbeing, second only to Japan (Varkey Foundation in the Guardian, 2017) in an international survey of 20 countries. Linked to this, more UK children than ever, 1 in 10, are suffering from mental health issues (NHS Digital, 2017; (Children's Society, 2008), yet services have diminished. Two thirds of those referred for specialist care received no treatment at all in 2017 (Spurgeons children's charity). At the same time, the number of children excluded from school continues to rise - there are now the equivalent of more than 35 permanent exclusions every school day in England (DfE, 2018). Persistent disruptive behaviour remains the most common reason for these exclusions (DfE, 2018) and we know that in the vast majority of cases, this behaviour is a cry for help and a signal of poor social and emotional wellbeing. We also know that excluded young people are more likely to end up in the criminal justice system. Around 60% of the prison population were excluded from school (IPPR). Pupils excluded by the age of 12 are four times more likely to be jailed as adults (McAra, L. & McVie, S, 2010). The UK prison system is struggling to cope with increasing levels of violence and

assault and the proven reoffending rate is unacceptably high for juvenile offenders at over 40% (Ministry of Justice, 2018).

The majority of young people in custody, or at risk of entering custody, have experienced neglect, abuse and trauma. They often have a history of adverse childhood experiences, exclusion, and disempowerment. As many as 90% of people in prison are estimated to have mental health problems, (Durcan, 2016), and almost half the children in Young Offender Institutions are Looked After Children (Prison Reform Trust, 2018). Childhood years are vital for developing positive social and emotional skills and well-being. Traumatic or adverse experiences in the crucial early years have a damaging effect on the development of these core cognitive and emotional skills, which are essential for managing thoughts, feelings, and behaviour, as well as interactions with others (WHO, 2012).

Many of the young people who come into contact with the criminal justice system carry a deep sense of shame and have been negatively labelled and excluded from society. Identity loss, low self-esteem and a socially devalued sense of self are all markers of poor mental well-being (Thoits in Sharma & Sharma) and also a central driver of criminal behaviour (Maruna and Farrall, 2004; McNeill and Weaver, 2010 in Beyond Youth Custody).

**Our Participants:** We believe that all young people should have access to quality SEL, however we focus our limited resources on providing this for young people who are most at risk of exclusion, offending or re-offending. Khulisa works with young people who:

- Suffer from poor mental health and low levels of social and emotional well-being;
- Have experienced trauma and / or adverse childhood experiences;
- May have behaved violently (physically or non-physically) towards themselves or others;
- Have been or are at risk of being excluded, marginalised and labelled;
- Lack confidence, self-esteem, self-worth and a sense of identity;

All of our young participants have potential and courage. We work with these young people because we believe that change is possible. We understand the effects of trauma and adverse childhood experiences and how they present in the body and are expressed through behaviour. We have identified an unmet need to treat young people who've been excluded from school or society with respect, and to work with them as the central agents of their own journey to positive change.

#### How do we work?

The Khulisa programme is **emergent and participant centered**. Khulisa's therapeutically-trained facilitators work through the content that is most relevant for the needs of the specific participants in the room, at a pace that matches their ability to absorb the learning. This means that no Khulisa programme is exactly the same as another.

We deliver the programme through a mixture of group activities and individual reflection sessions, using a range of creative activities including storytelling, mask-making, games and role-play. The programme is delivered by qualified art and drama therapists who use a therapeutic process to support the young people through a journey of self-awareness, self-discovery and realisation.

The programme is based on evidence of what works to build key social and emotional skills and is centered around 5 core approaches:

**Dramatherapy**: Khulisa's trained art and drama therapists use creative techniques (e.g. music, art, role-play, story-telling). These activities are associated with increased self-esteem, self-efficacy, empowerment, social and emotional competency, emotional intelligence and resilience (Daykin, 2008; Bungay, 2013, Zarobe and Bungay 2017).

**Small Group and 1-1 sessions**: Our peer groups explore positive and negative relationships together, while our ongoing 1-1 sessions help to embed individual learning. This approach is proven to develop emotional intelligence and social and emotional competence (Clarke, 2015).

**Asset-based theory:** through appreciation circles and strength-based observation, we help children realise and build on their strengths, essential in developing confidence and coping skills. This is proven to be particularly effective in reducing anxiety, improving coping skills and resilience (Collins, 2004; Sin et al., 2009; Neil et al. 2009).

**Restorative Approaches:** techniques such as circle dialogs, talking pieces, sociograms etc. empower young people to improve their social and emotional competency, relationships and emotional intelligence (Ortega et al., 2016).

#### **The Process of Change**

#### **Short-term Changes**

A range of evidence and direct delivery experience, supports the importance of the six clusters of social and emotional skills outlined below for social and emotional well-being and positive longer-term life outcomes (Young Foundation, 2012, Education Endowment Foundation, 2017). These competencies are **inter-connected and at times overlapping**. Although the programme is designed to develop this broad spectrum of social and emotional skills, **improved resilience**, **coping skills and emotional self regulation are prioritised as key short-term outcomes**.

These skills are the main focus of the programme and are seen as providing the foundation for the successful development of other social and emotional skills. This relates to Dr Bruce Perry's 'The

Three R's' model (Regulate, Relate, Reason) for learning among young people who have experienced trauma (Dr Bruce Perry, Three Rs Model). Heading straight for the 'Reasoning' part of the brain is unlikely to be successful if the young person is dysregulated and disconnected from others. First we must help the child to regulate and calm their flight / fight / freeze responses. Second, we must build trust, relate and connect. We must build resilience and coping skills to lay the foundation for the young person to engage with more challenging parts of the programme. Only then can we effectively support the young person to learn, reason, reflect, articulate, remember and become self-assured enough to fully engage.



#### **Longer-term Changes**

Improved social and emotional skills form the basis for improved longer-term social and emotional wellbeing, and positive life outcomes. These longer-term outcomes are not limited to the absence of crime, exclusion or negative behaviour. They include meaningful engagement with others and society, positive and productive life choices and a lifestyle that promotes well-being (Goodfellow et al, 2015 in BYC). In practice, this will look different for every individual. The focus is on flourishing and thriving rather than compliance and desistance.

Overall, we look for positive long-term changes in the following outcomes across all programmes:

• Social and emotional wellbeing – we measure both how a participant feels and how well they feel they are functioning - this is the key to achieving positive longer-term outcomes.

Depending on the type of intervention delivered, we also monitor the following longer-term observable behaviours:

- In-school / prison behaviour
- Academic attainment
- Return to mainstream schooling
- Re-offending rates
- Engagement in productive activity
- Transition to independent living
- Building strong support networks

Our own data shows that improved and social emotional skills and wellbeing are associated with positive external changes in behaviour. We believe that this positive behaviour in-turn further strengthens and reinforces wellbeing, promoting a positive and continued cycle of change over time. This process of change is complex and non-linear. Working with young people in difficult situations with complex needs requires intensive intervention and an awareness that relapse is possible as part of this process.

#### Khulisa's Theory of Change Diagram

The below image brings together short and longer-term outcomes, illustrating Khulisa's overall high-level Theory of Change:



#### **Enabling Factors:**

Listed below are the key enabling factors that we believe need to be in place for the intervention to be successful:

- Highly skilled, trauma-informed drama-therapists are adept at working with young people;
- Positive relationships and a sense of trust between the Khulisa facilitator(s), and with the other group members;
- Khulisa facilitators self-disclose, creating an open, safe environment;

- Young people feel respected and feel no judgement throughout the programme;
- Young people feel a sense of enjoyment, fulfilment and / or achievement as part of the programme;
- Young people feel that their voice is heard throughout the programme;
- Carefully selected partner institutions (schools pupil referral units, prisons, community organisations) share our core values and vision of success;
- Partner institutions understand the power of monitoring and evaluation and support and engage with data collection activities;
- Professionals in partner institutions are willing to fully engage with and adopt the Khulisa methodology;
- A prison and education sector that is able to invest in preventative solutions for the long-term.

#### **Our Assumptions**

While there is strong, consistent evidence proving the importance of social and emotional skills and wellbeing for positive life outcomes, specific evidence around what works and the causal mechanisms of change is still emerging. For this reason, we recognise that the intervention is based on a series of assumptions.

#### Causal link assumptions:

- Overall social and emotional wellbeing is strongly influenced by the 6 clusters of social and emotional skills identified in the framework presented above (the EEF SPECTRUM framework), in particular, resilience and coping;
- Improvements in social and emotional wellbeing resulting from Khulisa's intervention are sustained over the long-term (at least 12 months post intervention);
- Positive social and emotional wellbeing promotes positive mental health;
- Improved knowledge, skills and wellbeing of professionals leads to improvements in the social and emotional skills and wellbeing of the young people they support.

Equally important for the success of the programme are a series of practical implementation-focused assumptions:

- Partner institutions are selected purposefully and rigorously to ensure mutual responsibility for programme success;
- Partner institutions share the same values and vision;
- Partner institutions have the resources, commitment, leadership and capacity to translate trauma-informed theory into practice;
- Partner institutions fully understand and buy-in to the Khulisa methodology;
- The availability of a consistent, private, safe and adequate room in which programme delivery can take place without disruption;
- The ability of Khulisa facilitators to create a space where participants feel calm and able to openly express themselves without fear of judgement.

 Participants are able to commit to the process and are able to show up for the programme consistently.

#### What Makes Khulisa Unique?

Khulisa is providing a service that is currently not available for young people in schools, prisons and community organisations across the UK. We are the only organisation to provide all of the following as part of one package:

- Intensive support to young people most at need, addressing root causes not symptoms;
- Targeted support for young people with complex needs;
- A whole school / prison approach, aspiring to create cultural change and embedding our services in an institution over a significant period of time (usually 3 years) until sustainable institutional-level change is achieved;
- Programmes run only by **highly qualified art and drama therapists** who are skilled enough to deliver our methodology via a flexible approach whilst guaranteeing safety and security;
- Methodology built on an strengths-based approach (incorporating the Good Lives Model) recognising the assets and abilities of the young people we work with, no matter what situation they are in;
- A strong commitment to evidence-based approaches with commitment to quality monitoring and evaluation to use data to influence policy as well as practice.

#### References

- Beyond Youth Custody: Supporting the Shift: Framework for the effective resettlement of young people leaving custody accessed: http://www.beyondyouthcustody.net/wp-content/uploads/Now-all-I-care-about-is-my-futur e-Supporting-the-shift-full-research-report.pdf
- Bungay, H. & Vella-Burrows, T., "The Effects of Participating in Creative Activities on the Health and Well-Being of Children and Young People: A Rapid Review of the Literature." Vol.133 (1) (2013) Perspectives in Public Health pp44-52
- Education Endowment Foundation; (2017) Social, Psychological, Emotional, Concepts of self, and Resilience outcomes: Understanding and Measurement (SPECTRUM) A brief report of a conceptual mapping exercise accessed: https://educationendowmentfoundation.org.uk/public/files/Evaluation/SPECTRUM/EEF\_SPE
  - https://educationendowmentfoundation.org.uk/public/files/Evaluation/SPECTRUM/EEF\_SPE CTRUM\_Guidance\_Document\_Conceptual\_mapping.pdf
- World Health Organisation (2012), Risks to Mental Health: An Overview of Vulnerabilities and Risk Factors
  - http://www.who.int/mental\_health/mhgap/risks\_to\_mental\_health\_EN\_27\_08\_12.pdf
- Sharma, S. & Sharma, M. Psychol Stud (2010) 55: 118. https://doi.org/10.1007/s12646-010-0011-
- Cefai, C.; Bartolo P. A.; Cavioni. V; Downes, P.; Strengthening Social and Emotional Education as a core curricular area across the EU. A review of the international evidence, NESET II report, Luxembourg: Publications Office of the European Union, 2018. doi: 10.2766/664439
- The Young Foundation (2012), A framework of outcomes for young people accessed:
   https://assets.publishing.service.gov.uk/government/uploads/system/uploads/attachment\_d
   ata/file/175476/Framework\_of\_Outcomes\_for\_Young\_People.pdf

- Young Minds, 2006, accessed: https://youngminds.org.uk/search-results/?terms=mental+health+and+wellbeing
- Huppert FAaBN (2004) Well-being: towards an integration of psychology, neurobiology and social science. Biological Sciences 358 1447.
- Ryff CD, B. H. Singer, et al. (2004) Positive health: connecting well-being with biology. Philosophical Transactions of the Royal Society B: Biological Sciences 359: 1383.
- Keyes C.L.M. (2007) Promoting and protecting mental health as flourishing: A complementary strategy for improving national mental health. American Psychologist 62: 95.
- Steptoe A WJ, Marmot M. (2005) Positive affect and health-related neuroendocrine, cardiovascular, and inflammatory processes. Proceedings of the National Academy of Sciences of the United States of America 102: 6508.
- Chida Y SA (2008) Positive psychological well-being and mortality: A quantitative review of prospective observational studies. Psychosomatic Medicine 70: 741.
- McAra, L. & McVie, S, 2010). Youth Crime and Justice: Key Messages from the Edinburgh Study of Youth Transitions and Crime. Criminology & Criminal Justice, Vol.10(2), pp.179-209
- Ministry of Justice, "Her Majesty's Prison and Probation Service Offender Equalities Annual Report 2017/18" (2018)
- Durcan, G. (2016). Mental health and criminal justice: Views from consultations across
   England and Wales. Centre for Mental Health
- Prison Reform Trust, "Prison: The Facts" Bromley Briefings (2018)
- Zarobe, L and Bungay, H "The role of arts activities in developing resilience and mental wellbeing in children and young people a rapid review of the literature" Vol.137 (6) (2017) Perspectives in Public Health pp337-347

#### Annex C: Power calculations

Power calculations using a within-schools design can be found below.

| Within-schools trial | | |
|----------------------|-------------|------|
| n | n (per arm) | MDES |
| 160 | 80 | 0.45 |

Power calculation was determined on the basis the following assumptions:

• Power: 0.8

• Significance level: 0.05

• Level of randomisation: individual-level (i.e. individual students will be randomised)

• Number of trial arms: 2 (i.e. intervention and control)

• Outcome measure: SDQ

• Standard deviation: 6.5 in both groups

#### Stata code:

power twomeans 10, n(160) power(0.5) sd(6.5)

#### Annex D: Face It milestones

The following activities have been identified by Khulisa as essential to the core content of the Face It intervention. As such, while elements of programme content may vary in timing and specific implementation, a programme must contain all of these activities to be considered to be a typical Face It intervention.

The following activities comprise the 5-day programme; core activities are highlighted in bold.

| Day 1 | Intro and contracting | Recap why we are here |
|---|---|---|
| | | Recap what the programme is and how it will work |
| | | Icebreaker |
| | | Check-in circle |
| | | Code of honour |
| | | Check-out |
| | Understanding me | Check-in circle |
| | | Game |
| | | There's a hole in my pavement |
| | | Sociograms |
| | | Game |
| | | Check-out |
| | Introduction to triggers | Check-in circle |
| | | Game |
| | | Recap AM session |
| | | Cookie story |
| | | Window of tolerance |
| | | Emotional literacy wall/mapping |

| | | Game |
|-------|----------------------|----------------------------|
| | | Check-out |
| Day 2 | Triggers continued | Check-in |
| | | Game |
| | | Recap |
| | | Trigger game |
| | | Triggers |
| | | Game |
| | | Check-out |
| | Emotional literacy | Check-in |
| | | Game |
| | | Fight, flight, freeze |
| | | Body mapping |
| | | Intro to brain development |
| | | Game |
| | | Check-out |
| | Embedding emotional | Check-in |
| | literacy | Game |
| | | Iceberg |
| | | Grounding activity |
| | | Game |
| | | Check-out |
| Day 3 | Exploring challenges | Check-in |
| | | Game |
| | | Recap |
| | | Sociograms |
| | | Step in the middle |

| | | The 3 levels of violence |
|---|---|---|
| | | Game |
| | | Check-out |
| | Challenges continued | Check-in |
| | | Game |
| | | Role play |
| | | Inferior/superior |
| | | Game |
| | | Check-out |
| | Challenge cycle | Check-in |
| | | Game |
| | | Challenge cycle |
| | | Embedding learning |
| | | Game |
| | | Check-out |
| Day 4 | Understanding impact | Check-in |
| | of behaviour and developing coping | Game |
| | skills | Ripple effect |
| | | Are you a carrot, egg, or coffee bean |
| | | Coping skills activity |
| | | Embedding coping skills |
| | | Game |
| | | Check-out |
| | Accepting my mask | Check-in |
| | | Game |
| | | Please hear what I am not saying |
| | | Mask-making |

| | | Check-out |
|-------|-----------------------|---------------------------------|
| | Accept and appreciate | Check-in |
| | me | Game |
| | | Poem |
| | | Hat-making |
| | | Game |
| | | Check-out |
| Day 5 | Asset building | Check-in |
| | | Game |
| | | Recap |
| | | 3rd person intro |
| | | Game |
| | | Check-out |
| | Future focus | Check-in |
| | | Game |
| | | Future/back |
| | | Dragon's den |
| | | Two wolves: A Cherokee Teaching |
| | | Game |
| | | Check-out |
| | Appreciation and | Check-in |
| close | ciose | Game |
| | | Sweet appreciation |
| | | Pencil-maker |
| | | Game |
| | | Check-out |

## Annex E: Evaluation team experience

- Tom McBride is the Director of the Ending Youth Violence Lab and has over 15
  years of experience in research and evaluation roles. He is the former Director of
  Evidence at the Early Intervention Foundation and Head of Strategic Analysis at the
  Department for Education. Tom will have overall responsibility for the delivery and
  quality of this work.
- Jack Martin is an Assistant Director within the Ending Youth Violence Lab and has over 8 years of experience working at the Early Intervention Foundation and sits on the Government's Trials Advice Panel. Jack will oversee the delivery of the work and support, supervise and quality assure the work of the project team.
- Alice Worsley is an Associate Policy Advisor based in the Health and Wellbeing team at BIT. She has worked on projects across a range of policy areas and methodologies. Alice will project manage and coordinate the project.
- Patrick Taylor is a Principal Research Advisor and leads BIT's education and youth evaluation work, supporting the design, improvement and evaluation of complex interventions in these fields. Patrick will provide support and quality assurance for the pilot evaluation.
- Naomi Jones is a highly experienced social research consultant who specialises in helping organisations to design, commission, deliver and use research better, with over 18 years applied research experience. Naomi was formerly head of social attitudes at NatCen, where she led a mixed-method research team and oversaw the British Social Attitudes Survey. Naomi will lead the qualitative evaluation.
- Lilli Wagstaff is a quantitative research advisor in the Home Affairs and Security team at BIT and leads the evaluation and day-to-day delivery of a number of projects focusing on policy areas including reducing violence and recidivism. Lilli will lead the quantitative evaluation.
- Niall Daly is a Research Advisor in the Health and Wellbeing team at BIT, specialising in trial design, implementation, and quantitative data analysis across a range of projects within the health space. He will support the quantitative evaluation.
- Tess Moseley-Roberts is an Associate Policy Advisor in the Home Affairs, Security
  and International Development team at BIT. She has worked across peacebuilding,
  anti-corruption and education in the international space and a number of UK criminal
  justice projects. Tess will support the qualitative evaluation.

 Dr Nick Axford is an Associate Professor at the University of Plymouth with a specialism in evidence-based prevention and early intervention to improve child well-being, with a particular focus on developing or adapting interventions and evaluating their effectiveness and implementation. Nick has been a Member of the Early Intervention Foundation Evidence Panel since 2014 and will be providing expert advice and challenge on the design and delivery of the evaluation on a consultancy basis.

## Annex F: Schedule for recruitment, interventions and assessments

| Procedures | Data collection timepoints | | | | |
|---|---|---|---|---|---|
| | Screening | Baseline | Treatment phase | End-of-programme | 3-month follow-up |
| Referral form | | | | | |
| Screening log | | l | | | |
| Eligibility | | l | | | |
| Informed consent | | | | | |
| Demographics | | l | | | |
| Randomisation | | | | | |
| Intervention delivery | | | | | |
| Compliance | | | | | |
| Fidelity measures | Screening | Baseline | Treatment phase | End-of-programme | 3-month follow-up |
| Attendance/ engagement logs | | | | | |
| Session summary forms | | | | | |
| Outcome measures | Screening | Baseline | Treatment phase | End-of-programme | 3-month follow-up |

| School attendance |
|---|
| SDQ (parent and young person self-assessment) |
| SWEMWBS |
| Children's Hope Scale |
| The Emotional Regulation Questionnaire |
| The Self-Report Delinquency Scale |
| The Problem Behaviour Frequency Scale (overt and relational victimisation subscales only) |
| School Exclusion |
| Acceptability of content |
| Control group services as usual received |
| Qualitative interviews with young people |
| Qualitative interviews with parents |

| Qualitative interviews with key school staff |
|----------------------------------------------|
| Qualitative interviews with practitioners |
| Withdrawal from programme |

## Annex G: BIT data protection policy summary

The General Data Protection Regulation (GDPR) imposes certain obligations upon Behavioural Insights Limited (BIT), and other companies within the group, as Controllers and / or Processors in relation to processing Personal Data.

BIT takes these obligations seriously. BIT is committed to respecting the rights of all individuals whose personal data it processes:

- In relation to data security. BIT has implemented appropriate measures to ensure
  the secure storage and handling of Personal Data, including obtaining a Cyber
  Essentials Plus certification and developing a comprehensive Data Handling
  Protocol.
- 2. In relation to data protection and privacy rights, our data processing activities are conducted according to the principles relating to the processing of Personal Data set out in the GDPR, including that Personal Data shall be processed lawfully, fairly and in a transparent manner, and in a manner that ensures the security of the Personal Data. BIT has policies and procedures in place to ensure compliance with these principles.

More information on how we handle Personal Data in relation to projects we are working on is detailed below.

BIT is registered with the UK ICO under the terms of the Data Protection Act 2018. Our registration number is ZA038649.

#### Privacy by design

BIT conducts all trials and research projects with a privacy by design approach to protect and maintain the privacy and security of research participants' and research subjects' data. We work closely with clients, government departments and research partners when designing interventions to ensure that a privacy by design approach is implemented and respected.

Our data protection and data security policies and procedures reflect necessary legislative requirements and set out the standard to which BIT staff should work when dealing with Personal Data, including:

- Attendance at mandatory data protection training for all employees;
- Identifying data requirements from the outset of each project;
- Minimising use of Personal Data where possible and ensuring we have the right to handle any Personal Data where successful project delivery is reliant on using it;
- Putting in place data processing agreements with all clients and suppliers to clarify data handling arrangements ahead of any data being transferred;

- Complying with all relevant data residency requirements and implementing appropriate technical and organisational measures, to protect data and avoid unauthorised access, internally and externally;
- A clear internal reporting process in the event of a data breach, to consider the
  nature of the breach and identify any necessary action, including whether the breach
  should be reported to the relevant authorities, i.e. the Information Commissioner's
  Office in the UK or the Office of the Australian Information Commissioner;
- Clear procedures on retention and destruction of Personal Data to avoid keeping hold of Personal Data longer than necessary for the purposes of each project; and
- Implementing robust investigation and reporting procedures in relation to any data breach or security issues that arise both within our own systems and those of our clients, partners and suppliers.

#### **Data Protection Officer**

The BIT group of companies has appointed a Data Protection Officer (DPO) who is the first point of contact for any issue regarding data protection and data security. The DPO can be contacted via email at legal@bi.team or by writing to us at:

Legal Team, Behavioural Insights Limited, 58 Victoria Embankment, London, EC4Y 0DS, United Kingdom.